CLINICAL TRIAL: NCT04886596
Title: A Phase 3, Randomized, Placebo-controlled, Observer-blind, Multi-country Study to Demonstrate the Efficacy of a Single Dose and Annual Revaccination Doses of GSK's RSVPreF3 OA Investigational Vaccine in Adults Aged 60 Years and Above
Brief Title: Efficacy Study of GSK's Investigational Respiratory Syncytial Virus (RSV) Vaccine in Adults Aged 60 Years and Above
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 212494; 2020-000753-28 (EudraCT Number)
Record Dates: First submitted 2021-04-29; First posted 2021-05-14 (Actual); Results first posted 2023-08-04 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory syncytial virus; Lower respiratory tract disease; Efficacy study; Adults aged 60 years and above
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is an observer blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RSVPreF3 Group (Experimental): Participants received a single dose of the RSVPreF3 OA vaccine at Day 1. Before the second vaccination participants in this group were re-randomized into 2 as: a group that received placebo every subsequent year, and a group that received an additional dose of RSVPreF3 OA vaccine every subsequent year of the study.
  Interventions: Biological: RSVPreF3 OA vaccine
- Placebo Group (Placebo Comparator): Participants received 1 dose of placebo at Day 1 and an additional dose of placebo every subsequent year of the study.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Placebo — Placebo administered intramuscularly into the deltoid of the non-dominant arm at day 1 and before Season 2 to the Placebo Group, and before Season 2 to the participants of the RSVPreF3 Group, that are re-randomized to the RSV_1 dose group.
  Arms: Placebo Group
Biological: RSVPreF3 OA vaccine — RSVPreF3 OA vaccine administered intramuscularly into the deltoid of the non-dominant arm at Day 1 in the RSVPreF3 group, and before Season 2 to the participants of the RSVPreF3 group that are re-randomized to the RSV_annual group.
  Arms: RSVPreF3 Group

SUMMARY:
This study will evaluate the efficacy of the RSVPreF3 OA investigational vaccine in preventing Lower Respiratory Tract Disease (LRTD) caused by RSV in adults ≥60 years of age following a single dose of the RSVPreF3 OA vaccine and following annual revaccination doses in Northern Hemisphere (NH) and in Southern Hemisphere (SH). This study will also assess if the vaccine is safe and induces an immune response.

DETAILED DESCRIPTION:
Dose 1 Period will be conducted in 2 parts: Part 1: Participants in RSVPreF3 groups will receive lots 1, 2 and 3 of the investigational vaccine before Season 1. Part 2: Will be initiated when the vaccine lots in part 1 are exhausted at the study sites and participants in RSVPreF3 group will receive lot 4 of the investigational vaccine before Season 1.

ELIGIBILITY:
Inclusion Criteria:

* A male or female ≥ 60 YOA at the time of first vaccination, who live in the community (community dwelling participants) or in a long-term care facility (LTCF participants).
* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol.

Note: In case of physical incapacity that would preclude the self-completion of the diary cards and/or questionnaires, either site staff can assist the participant (for activities performed during site visits) or the participant may assign a caregiver to assist him/her with this activity (for activities performed at home or in the LTCF). However, at no time, the site staff or caregiver will evaluate the participant's health status while answering diaries and/or questionnaires or make decisions on behalf of the participant

* Written or witnessed informed consent obtained from the participant prior to performance of any study specific procedure.
* Participants who are medically stable in the opinion of the investigator at the time of first vaccination. Participants with chronic stable medical conditions with or without specific treatment, such as diabetes, hypertension or cardiac disease, are allowed to participate in this study if considered by the investigator as medically stable.

Exclusion Criteria:

Medical conditions

* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease or immunosuppressive/cytotoxic therapy, based on medical history and physical examination (no laboratory testing required).
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Hypersensitivity to latex.
* Serious or unstable chronic illness.
* Any history of dementia or any medical condition that moderately or severely impairs cognition.

Note: If deemed necessary for clinical evaluation, the investigator can use tools such as Mini-Mental State Exam (MMSE), Mini-Cog or Montreal Cognitive Assessment (MoCA) to determine cognition levels of the participant.

* Recurrent or un-controlled neurological disorders or seizures. Participants with medically-controlled active neurological diseases can be enrolled in the study as per investigator assessment, provided that their condition will allow them to comply with the requirements of the protocol.
* Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.

Prior/Concomitant therapy

* Use of any investigational or non-registered product (drug, vaccine or medical device) other than the study vaccine during the period beginning 30 days before the first study vaccine administration, or planned use during the study period.
* Planned or actual administration of a vaccine not foreseen by the study protocol in the period starting 30 days before each dose and ending 30 days after each dose of study vaccine administration, with the exception of inactivated and subunit influenza vaccines which can be administered up to 14 days before or from 14 days after each study vaccination.
* Previous vaccination with an RSV vaccine.
* Administration of long-acting immune-modifying drugs or planned administration at any time during the study period.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 90 days before the first study vaccine or planned administration during the study period.
* Chronic administration (defined as more than 14 consecutive days in total) of immunosuppressants or other immune-modifying drugs during the period starting 90 days prior to the first study vaccine administration or planned administration during the study period. For corticosteroids, this will mean prednisone ≥20 mg/day, or equivalent. Inhaled and topical steroids are allowed.

Prior/Concurrent clinical study experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product (drug or medical device).

Other exclusions

* History of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential participant unable/unlikely to provide accurate safety reports or comply with study procedures.
* Bedridden participants.
* Planned move during the study period that will prohibit participating in the trial until study end. This includes:

  * Planned move during the study period to another LTCF that will prohibit participation in the trial until study end.
  * Planned move from the community to a LTCF that will prohibit participation in the trial until study end.
* Participation of any study personnel or their immediate dependants, family, or household members.
* Planned leave or holiday of 4 consecutive weeks or more during the RSV seasons* covered by the study, that would prohibit the reporting of ARI cases and attendance to ARI visit.

  * RSV seasons are from October to April in NH and from March to September in SH.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26675 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (228):
- United States (57):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Cerritos, California
  - GSK Investigational Site, Laguna Hills, California
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Lake City, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Pinellas Park, Florida
  - GSK Investigational Site, The Villages, Florida
  - GSK Investigational Site, Weeki Wachee, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Mishawaka, Indiana
  - GSK Investigational Site, El Dorado, Kansas
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Richfield, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Binghamton, New York
  - GSK Investigational Site, Jamaica, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Rocky Mount, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Statesville, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Centerville, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Keller, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Norfolk, Virginia
- Australia (9):
  - GSK Investigational Site, Botany, New South Wales
  - GSK Investigational Site, Coffs Harbour, New South Wales
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Morayfield, Queensland
  - GSK Investigational Site, Taringa, Queensland
  - GSK Investigational Site, Tarragindi, Queensland
  - GSK Investigational Site, Camberwell, Victoria
  - GSK Investigational Site, Geelong, Victoria
  - GSK Investigational Site, Spearwood, Western Australia
- Belgium (10):
  - GSK Investigational Site, Aalst
  - GSK Investigational Site, Alken
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Erpent
  - GSK Investigational Site, Genk
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Ieper
  - GSK Investigational Site, Linkebeek
  - GSK Investigational Site, Mechelen
  - GSK Investigational Site, Tremelo
- Canada (19):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, New Westminster, British Columbia
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, London-Ontario, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Sarnia, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Chicoutimi, Quebec
  - GSK Investigational Site, Mirabel, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Estonia (3):
  - GSK Investigational Site, Paide
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Finland (9):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- Germany (22):
  - GSK Investigational Site, Freiberg, Saxony
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Cologne
  - GSK Investigational Site, Dachau
  - GSK Investigational Site, Dippoldiswalde
  - GSK Investigational Site, Dresden
  - GSK Investigational Site, Essen
  - GSK Investigational Site, Flörsheim
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Freital
  - GSK Investigational Site, Goch
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Hanover
  - GSK Investigational Site, Leipzig
  - GSK Investigational Site, Mainz
  - GSK Investigational Site, München
  - GSK Investigational Site, Schenefeld
  - GSK Investigational Site, Wallerfing
  - GSK Investigational Site, Wangen
  - GSK Investigational Site, Weinheim
  - GSK Investigational Site, Witten
  - GSK Investigational Site, Würzburg
- Italy (15):
  - GSK Investigational Site, Alessandria
  - GSK Investigational Site, Bari
  - GSK Investigational Site, Belluno
  - GSK Investigational Site, Catanzaro
  - GSK Investigational Site, Chieri Torino
  - GSK Investigational Site, Ferrara
  - GSK Investigational Site, Genova
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Napoli
  - GSK Investigational Site, Negrar Verona
  - GSK Investigational Site, Palermo
  - GSK Investigational Site, Pisa
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Siena
  - GSK Investigational Site, Vercelli
- Japan (11):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Okinawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Yamagata
  - GSK Investigational Site, Yamaguchi
- Mexico (9):
  - GSK Investigational Site, Chihuahua City
  - GSK Investigational Site, León
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, Mérida
  - GSK Investigational Site, Monterrey
  - GSK Investigational Site, Oaxaca City
  - GSK Investigational Site, Querétaro
  - GSK Investigational Site, RM Pharmamexico CITY
  - GSK Investigational Site, San Luis Potosí City
- New Zealand (6):
  - GSK Investigational Site, Grafton Auckland
  - GSK Investigational Site, Havelock North
  - GSK Investigational Site, Kapiti
  - GSK Investigational Site, Palmerston North
  - GSK Investigational Site, Tauranga
  - GSK Investigational Site, Wellington
- Poland (11):
  - GSK Investigational Site, Częstochowa
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Gdynia
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Piaseczno
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Russia (7):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Gatchina
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, StPetersburg
  - GSK Investigational Site, Yekaterinburg
- South Africa (7):
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, Middelburg
  - GSK Investigational Site, Moloto South
  - GSK Investigational Site, Newcastle
  - GSK Investigational Site, Reiger Park
  - GSK Investigational Site, Tembisa
- South Korea (8):
  - GSK Investigational Site, Ansan
  - GSK Investigational Site, Bucheon-si Kyunggi-do 14584
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Jeonju
  - GSK Investigational Site, Kangwon-do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon Gyeonggi-do
- Spain (5):
  - GSK Investigational Site, Alcorcón
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Valencia
- United Kingdom (20):
  - GSK Investigational Site, Bebington
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Bradford on Avon Wiltsh
  - GSK Investigational Site, Cardiff
  - GSK Investigational Site, Corby
  - GSK Investigational Site, Eynsham
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Hardwick
  - GSK Investigational Site, Hexham
  - GSK Investigational Site, Lancashire
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Orpington
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Peterborough
  - GSK Investigational Site, Romford
  - GSK Investigational Site, Royal Leamington Spa
  - GSK Investigational Site, Thetford Norfolk
  - GSK Investigational Site, Witney

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer tohttps://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

REFERENCES:
- [Background] Ison MG, Papi A, Athan E, Feldman RG, Langley JM, Lee DG, Leroux-Roels I, Martinon-Torres F, Schwarz TF, van Zyl-Smit RN, Verheust C, Dezutter N, Gruselle O, Fissette L, David MP, Kostanyan L, Hulstrom V, Olivier A, Van der Wielen M, Descamps D; AReSVi-006 Study Group. Efficacy and Safety of Respiratory Syncytial Virus (RSV) Prefusion F Protein Vaccine (RSVPreF3 OA) in Older Adults Over 2 RSV Seasons. Clin Infect Dis. 2024 Jun 14;78(6):1732-1744. doi: 10.1093/cid/ciae010. PMID 38253338
- [Derived] Tajima K, Zarkadoulas E, Simons J, Kurai D, Grace M, Graham J, Ho Y, Verelst F. Cost-effectiveness of the adjuvanted respiratory syncytial virus prefusion F protein (RSVPreF3) vaccine in Japanese adults aged 50-59 years at increased risk of severe RSV disease and those aged >/=60 years. Expert Rev Vaccines. 2026 Feb 4:2626921. doi: 10.1080/14760584.2026.2626921. Online ahead of print. PMID 41637686
- [Derived] Ison MG, Papi A, Athan E, Feldman RG, Langley JM, Lee DG, Leroux-Roels I, Martinon-Torres F, Schwarz TF, van Zyl-Smit RN, Cuadripani S, Deraedt Q, Dezutter N, Gerard C, Fissette L, Xavier S, David MP, Olivier A, Van der Wielen M, Descamps D; AReSVi-006 study group. Efficacy, safety, and immunogenicity of the AS01E-adjuvanted respiratory syncytial virus prefusion F protein vaccine (RSVPreF3 OA) in older adults over three respiratory syncytial virus seasons (AReSVi-006): a multicentre, randomised, observer-blinded, placebo-controlled, phase 3 trial. Lancet Respir Med. 2025 Jun;13(6):517-529. doi: 10.1016/S2213-2600(25)00048-7. Epub 2025 Apr 14. PMID 40245915
- [Derived] Sanchez-Martinez ZV, Alpuche-Lazcano SP, Stuible M, Durocher Y. CHO cells for virus-like particle and subunit vaccine manufacturing. Vaccine. 2024 Apr 11;42(10):2530-2542. doi: 10.1016/j.vaccine.2024.03.034. Epub 2024 Mar 19. PMID 38503664
- [Derived] Kurai D, Mizukami A, Preckler V, Verelst F, Molnar D, Matsuki T, Ho Y, Igarashi A. The potential public health impact of the respiratory syncytial virus prefusion F protein vaccine in people aged >/=60 years in Japan: results of a Markov model analysis. Expert Rev Vaccines. 2024 Jan-Dec;23(1):303-311. doi: 10.1080/14760584.2024.2323128. Epub 2024 Mar 1. PMID 38426479
- [Derived] Curran D, Matthews S, Cabrera ES, Perez SN, Breva LP, Ramet M, Helman L, Park DW, Schwarz TF, Melendez IMG, Schaefer A, Roy N, Stephan B, Molnar D, Kostanyan L, Powers JH 3rd, Hulstrom V; Members of the AReSVi-006 Study Group. The respiratory syncytial virus prefusion F protein vaccine attenuates the severity of respiratory syncytial virus-associated disease in breakthrough infections in adults >/=60 years of age. Influenza Other Respir Viruses. 2024 Feb 3;18(2):e13236. doi: 10.1111/irv.13236. eCollection 2024 Feb. PMID 38314063
- [Derived] Feldman RG, Antonelli-Incalzi R, Steenackers K, Lee DG, Papi A, Ison MG, Fissette L, David MP, Marechal C, Van der Wielen M, Kostanyan L, Hulstrom V; AReSVi-006 Study Group. Respiratory Syncytial Virus Prefusion F Protein Vaccine Is Efficacious in Older Adults With Underlying Medical Conditions. Clin Infect Dis. 2024 Jan 25;78(1):202-209. doi: 10.1093/cid/ciad471. PMID 37698366
- [Derived] Papi A, Ison MG, Langley JM, Lee DG, Leroux-Roels I, Martinon-Torres F, Schwarz TF, van Zyl-Smit RN, Campora L, Dezutter N, de Schrevel N, Fissette L, David MP, Van der Wielen M, Kostanyan L, Hulstrom V; AReSVi-006 Study Group. Respiratory Syncytial Virus Prefusion F Protein Vaccine in Older Adults. N Engl J Med. 2023 Feb 16;388(7):595-608. doi: 10.1056/NEJMoa2209604. PMID 36791160

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 26675 participants enrolled in the study, 24972 received study intervention and were included in the Exposed set and started the study.
Period: Overall Study
Arm/Group | RSVPreF3 Group | Placebo Group
Started | 12469 | 12503
RSV_1_dose (Participants that received placebo every subsequent year of the study after first dose of RSVPreF3 OA vaccine at Day 1.) | 6226 | 0
RSV_annual (Participants that received an adittional RSVPreF3 OA vaccine every subsequent year of the study after first dose of RSVPreF3 OA vaccine at Day 1.) | 6243 | 0
Completed | 9365 | 9361
Not Completed | 3104 | 3142
Not completed — Adverse Event | 442 | 441
Not completed — Lost to Follow-up | 448 | 465
Not completed — Consent withdrawal, not due to a (S)AE | 1715 | 1726
Not completed — Migrated/moved from the study area | 201 | 184
Not completed — Other | 298 | 326

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RSVPreF3 Group | Placebo Group | Total
Number analyzed (Participants) | 12469 | 12503 | 24972
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 69.5 (6.5) | 69.6 (6.4) | 69.5 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6489 | 6429 | 12918
  Male | 5980 | 6074 | 12054
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Races where 0<n<11 (i.e., Native Hawaiian or Other Pacific Islander and American Indian or Alaska Native) are combined into one category ("All Other Races") to maintain participant confidentiality and privacy.
  Participants
    Asian | 953 | 956 | 1909
    Black or African American | 1064 | 1101 | 2165
    White | 9889 | 9936 | 19825
    All Other Races | 55 | 41 | 96
    Other | 508 | 469 | 977

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Episode of RT-PCR Confirmed RSV A and/or B Associated Lower Respiratory Tract Disease (LRTD) During the First Season Following a Single Dose of the RSVPreF3 OA Vaccine
Description: First episode of Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR)-confirmed RSV A and/or RSV B- associated LRTD during the first season was assessed. The case definition for RSV-confirmed LRTD is as follows: Presence of at least one RSV-positive swab detected by RT-PCR.
Time Frame: From Day 15 post-vaccination up to end of season 1 in the Northern Hemisphere (NH) [a median of approximately 6.7 months (6.9 months in NH and 3.5 months in Southern Hemisphere [SH])]
Population: Analysis was performed on the modified Exposed Set (mES), which included all participants who received at least the first dose of the study intervention and who do not report an RSV-confirmed Acute Respiratory Illness (ARI) prior to 2 weeks (<Day 15) after each vaccination (mES-RSV set). Only participants with data available at specified timepoints were included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 12466 | 12494
Participants | 7 | 40
Statistical Analysis 1: Comparison: RSVPreF3 Group vs Placebo Group; To demonstrate the vaccine efficacy (VE) efficacy of a single dose of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD during the first season in adults ≥ 60 YOA; Test type: Other — VE is demonstrated if the lower limit (LL) of the 2-sided confidence interval (CI) for vaccine efficacy (VE) is above 20%; Poisson regression method; VE = 82.58, 96.95% CI 2-sided [57.89 to 94.08] — VE in terms of occurrence of RSV-confirmed LRTD was evaluated using the conditional exact binomial method based on the Poisson model

2. Secondary Outcome: Number of Participants With First Episode of RT-PCR Confirmed RSV A and/or B Associated LRTD Over Several Seasons Following a Single Dose of the RSVPreF3 OA Vaccine
Description: Efficacy of a single dose of the RSVPreF3 OA vaccine was assessed against RSV A and/or B confirmed LRTD over several seasons according to the case definition.
Time Frame: From Day 15 post first vaccination up to end of season 2 and up to end of season 3 in the Northern Hemisphere [NH] (assessed approximately over 2 and 3 years in NH)
Population: Analysis was performed on the mES-RSV. Only participants with data available at specified timepoints were included in analysis. For single dose evaluation, participants from the RSV_annual group who received RSVPreF3 OA investigational vaccine at Dose 2 contributed to Season 1 data only and were censored starting from Dose 2 administration.
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 12469 | 12498
Participants
  Season 2 (NH) | 30 | 139
  Season 3 (NH): number analyzed (Participants) | 12468 | 12498
  Season 3 (NH) | 48 | 215
Statistical Analysis 1: Comparison: RSVPreF3 Group vs Placebo Group; To demonstrate the vaccine efficacy of a single dose of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD in adults ≥ 60 YOA over three seasons; Test type: Other — VE is demonstrated if the LL of the 2-sided CI for VE is above 20%; Poisson regression method; VE = 62.91, 97.5% CI 2-sided [46.74 to 74.79] — VE is defined as 1 minus the relative risk (RR). RR=the ratio of the incidence rates of RSVPreF3 Group over Placebo Group. VE (%) = Vaccine Efficacy (Poisson method - adjusted by age, region and season)
Statistical Analysis 2: Comparison: RSVPreF3 Group vs Placebo Group; To demonstrate the vaccine efficacy of a single dose of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD in adults ≥ 60 YOA over two seasons; Test type: Other — VE is demonstrated if the LL of the 2-sided CI for VE is above 20%; Poisson regression method; VE = 67.18, 97.5% CI 2-sided [48.19 to 80.04] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Number of Participants With First Episode of RT-PCR Confirmed RSV A and/or B Associated LRTD Over Several Seasons Following Annual Revaccination Doses of the RSVPreF3 OA Vaccine
Description: Efficacy of annual revaccination doses of the RSVPreF3 OA vaccine was assessed against RSV A and/or B confirmed LRTD over several seasons according to the case definition.
Time Frame: From Day 15 post first vaccination up to end of season 2 and up to end of season 3 in the NH (assessed approximately over 2 and 3 years in NH)
Population: Analysis was performed on the mES-RSV. Only participants with data available at specified timepoints were included in analysis. For annual dose evaluation, participants from the RSV_1_dose group who received Placebo at Dose 2 contributed to Season 1 data only and were censored starting from Dose 2 administration.
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 12469 | 12498
Participants
  Season 2 (NH) | 30 | 139
  Season 3 (NH): number analyzed (Participants) | 12468 | 12498
  Season 3 (NH) | 38 | 192
Statistical Analysis 1: Comparison: RSVPreF3 Group vs Placebo Group; To demonstrate the vaccine efficacy of a single dose of the RSVPreF3 OA investigational vaccine followed by 1 annual revaccination before Season 2 in the prevention of RSV-confirmed LRTD in adults ≥ 60 YOA over three seasons; Test type: Other — VE is demonstrated if the LL of the 2-sided CI for VE is above 20%; Poisson regression method; VE = 67.76, 97.5% CI 2-sided [51.82 to 79.11] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: RSVPreF3 Group vs Placebo Group; To demonstrate the vaccine efficacy of a single dose of the RSVPreF3 OA investigational vaccine followed by 1 annual revaccination before Season 2 in the prevention of RSV-confirmed LRTD in adults ≥ 60 YOA over two seasons; Test type: Other — VE is demonstrated if the LL of the 2-sided CI for VE is above 20%; Poisson regression method; VE = 67.12, 97.5% CI 2-sided [48.09 to 80.00] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Number of Participants With First Episode of RT-PCR Confirmed RSV Subtype A and Subtype B LRTD Over 3 Seasons Following a Single Dose of the RSVPreF3 OA Vaccine
Description: Efficacy of a single dose of the RSVPreF3 OA vaccine was assessed against LRTD episode caused by RSV A and B subtype over 3 seasons according to the case definition.
Time Frame: From Day 15 post first vaccination up to end of season 3 in the NH (assessed approximately over 3 years in NH, and 2.5-3 years in SH)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 12468 | 12498
Participants
  RT-PCR-confirmed RSV-A LRTD | 14 | 80
  RT-PCR-confirmed RSV-B LRTD | 34 | 135
Statistical Analysis 1: Comparison: RSVPreF3 Group vs Placebo Group; To demonstrate the vaccine efficacy of a single dose of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD for RSV subtype A in adults ≥ 60 YOA over 3 seasons; Test type: Other — VE is demonstrated if the LL of the 2-sided CI for VE is above 0%; Poisson regression method; VE = 69.83, 97.5% CI 2-sided [42.18 to 85.72] — VE is defined as 1 minus the relative risk (RR). RR=the ratio of the incidence rates of RSVPreF3 Group over Placebo Group. VE (% ) = Vaccine Efficacy (Poisson method - adjusted by age, region and season)
Statistical Analysis 2: Comparison: RSVPreF3 Group vs Placebo Group; To demonstrate the vaccine efficacy of a single dose of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD for RSV subtype B in adults ≥ 60 YOA over 3 seasons; Test type: Other — VE is demonstrated if the LL of the 2-sided CI for VE is above 0%; Poisson regression method; VE = 58.57, 97.5% CI 2-sided [35.90 to 74.11] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Number of Participants With First Episode of RT-PCR Confirmed RSV Subtype A and Subtype B LRTD Over 3 Seasons Following a Single Dose of the RSVPreF3 OA Vaccine and Following 1 Annual Revaccination Dose
Description: Efficacy of a single dose and 1 annual revaccination dose of the RSVPreF3 OA vaccine was assessed against LRTD episode caused by RSV A and B subtype over 3 seasons according to the case definition.
Time Frame: as for outcome 4
Population: Analysis was performed on the mES-RSV. Only participants with data available at specified timepoints were included in analysis. For single dose evaluation, participants from the RSV_annual group who received RSVPreF3 OA investigational vaccine at Dose 2 contributed to Season 1 data only and were censored starting from Dose 2. For annual dose evaluation, participants from the RSV_1_dose group who received Placebo at Dose 2 contributed to Season 1 data only and were censored starting from Dose 2.
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 12468 | 12498
Participants
  RT-PCR-confirmed RSV-A LRTD | 17 | 65
  RT-PCR-confirmed RSV-B LRTD | 21 | 127
Statistical Analysis 1: Comparison: RSVPreF3 Group vs Placebo Group; To demonstrate the vaccine efficacy of a single dose and 1 annual revaccination before Season 2 of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD for RSV subtype A in adults ≥ 60 YOA over 3 seasons; Test type: Other — VE is demonstrated if the LL of the 2-sided CI for VE is above 0%; Poisson regression method; VE = 55.12, 97.5% CI 2-sided [16.52 to 77.52] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: RSVPreF3 Group vs Placebo Group; To demonstrate the vaccine efficacy of a single dose and 1 annual revaccination before Season 2 of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD for RSV subtype B in adults ≥ 60 YOA over 3 seasons; Test type: Other — VE is demonstrated if the LL of the 2-sided CI for VE is above 0%; Poisson regression method; VE = 73.58, 97.5% CI 2-sided [55.10 to 85.40] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Number of Participants With First Episode of RT-PCR Confirmed LRTD Caused by Human Metapneumovirus (hMPV) up to the End of Season 1 Following a Single Dose of the RSVPreF3 OA Vaccine
Time Frame: From Day 15 post-vaccination up to end of season 1 in the SH [a median of approximately 11.5 months (11.6 months in NH and 9.1 months in SH)]
Population: Analysis was performed on the mES-RSV. Only participants with data available at specified timepoints were included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 12469 | 12503
Participants | 53 | 65
Statistical Analysis 1: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of hMPV-confirmed LRTD in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine up to the end of Season 1; Test type: Other — The statistical analyses performed for the study objectives were descriptive. No success criteria were defined for the statistical analyses; Poisson regression method; VE = 18.41, 95% CI 2-sided [-19.10 to 44.33] — VE is defined as 1 minus the relative risk (RR). RR=the ratio of the incidence rates of RSVPreF3 Group over Placebo Group VE (% ) = Vaccine Efficacy (Poisson method - adjusted by age, region and season)

7. Secondary Outcome: Number of Participants With First Episode of RT-PCR Confirmed RSV A and/or B Associated LRTD, by Age Categories Following a Single Dose of the RSVPreF3 OA Vaccine and Following Annual Revaccination Doses
Description: Efficacy of a single dose of the RSVPreF3 OA vaccine and annual revaccination doses was assessed against RSV A and/or B confirmed LRTD episode according to the case definition, in the following age categories: greater than or equal to (≥) 65 years of age (YOA), ≥70 YOA and ≥80 YOA.
Time Frame: From Day 15 post first vaccination up to end of season 3 in the NH (assessed approximately over 3 years in NH and 2.5-3 years in SH)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 9261 | 9328
Participants
  RT-PCR-confirmed RSV LRTD (Single dose), >=65 YOA | 38 | 156
  RT-PCR-confirmed RSV LRTD (Single dose), >=70 YOA: number analyzed (Participants) | 5506 | 5517
  RT-PCR-confirmed RSV LRTD (Single dose), >=70 YOA | 20 | 98
  RT-PCR-confirmed RSV LRTD (Single dose), >=80 YOA,: number analyzed (Participants) | 1017 | 1028
  RT-PCR-confirmed RSV LRTD (Single dose), >=80 YOA, | 5 | 13
  RT-PCR-confirmed RSV LRTD (Annual revaccination), >=65 YOA | 28 | 137
  RT-PCR-confirmed RSV LRTD (Annual revaccination), >=70 YOA: number analyzed (Participants) | 5506 | 5517
  RT-PCR-confirmed RSV LRTD (Annual revaccination), >=70 YOA | 19 | 87
  RT-PCR-confirmed RSV LRTD (Annual revaccination), >=80 YOA: number analyzed (Participants) | 1017 | 1028
  RT-PCR-confirmed RSV LRTD (Annual revaccination), >=80 YOA | 5 | 12
Statistical Analysis 1: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD by >=65YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 58.78, 95% CI 2-sided [40.73 to 71.96] — VE is defined as 1 minus the relative risk (RR). RR=the ratio of the incidence rates of RSVPreF3 Group over Placebo Group. VE (% ) = Vaccine Efficacy (Poisson method - adjusted by region and season)
Statistical Analysis 2: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD by >=70YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 65.98, 95% CI 2-sided [44.32 to 80.16] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD by >=80YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 36.24, 95% CI 2-sided [-93.99 to 82.47] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD by >=65YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 66.56, 95% CI 2-sided [49.33 to 78.64] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 5: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD by >=70YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine at end of season 3; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 64.25, 95% CI 2-sided [40.49 to 79.55] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 6: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD by >=80YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine at end of season 3; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 32.81, 95% CI 2-sided [-108.42 to 81.73] — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Number of Participants With First Episode of RT-PCR Confirmed RSV A and/or B Associated LRTD by RSV Season Following a Single Dose of the RSVPreF3 OA Vaccine and Following Annual Revaccination Doses
Description: Efficacy of a single dose of the RSVPreF3 OA vaccine and annual revaccination doses was assessed against RSV A and/or B confirmed LRTD episode according to the case definition, by RSV season as follows: VE after each season includes the first occurrence of episodes reported from Day 15 post vaccination at first season, and for the next seasons, excluding analysis of participants who already reported a case in the previous season. The RSV season may be extended based on epidemiology data.
Time Frame: From Day 15 post first dose or start of the RSV season to the first occurrence of RSV-confirmed LRTD at each RSV season (assessed approximately over 7 months at each season [Seasons 1 and 2 in SH, Seasons 1, 2 and 3 in NH])
Population: Analysis was performed on the mES-RSV. Only participants with data available at specified timepoints were included in analysis. Analysis is presented based on the groups at each season (RSVPreF3 group for Season 1, RSV_1_dose and RSV_annual groups for Seasons 2 and 3, Placebo group for Season 1, 2 and 3).
Measure: Count of Participants; unit: Participants
Groups:
- RSV_1_dose Group: Participants received a dose of placebo every subsequent year after the vaccination at Day 1 of the study.
- RSV_annual Group: Participants received an additional dose of RSVPreF3 OA vaccine every subsequent year after the vaccination at Day 1 of the study.
Arm/Group | RSVPreF3 Group | Placebo Group | RSV_1_dose Group | RSV_annual Group
Number analyzed (Participants) | 12468 | 12498 | 4988 | 4968
Participants
  RT-PCR-confirmed RSV LRTD, Season 1: number analyzed (Participants) | 12468 | 12498 | 0 | 0
  RT-PCR-confirmed RSV LRTD, Season 1 | 7 | 36 |  |
  RT-PCR-confirmed RSV LRTD, Season 2 (Single dose): number analyzed (Participants) | 0 | 10031 | 4988 | 0
  RT-PCR-confirmed RSV LRTD, Season 2 (Single dose) |  | 98 | 19 |
  RT-PCR-confirmed RSV LRTD, Season 2 (Annual revaccination): number analyzed (Participants) | 0 | 10031 | 0 | 4968
  RT-PCR-confirmed RSV LRTD, Season 2 (Annual revaccination) |  | 98 |  | 22
  RT-PCR-confirmed RSV LRTD, Season 3 (Single dose): number analyzed (Participants) | 0 | 10031 | 4988 | 0
  RT-PCR-confirmed RSV LRTD, Season 3 (Single dose) |  | 60 | 16 |
  RT-PCR-confirmed RSV LRTD, Season 3 (Annual revaccination): number analyzed (Participants) | 0 | 7224 | 0 | 3582
  RT-PCR-confirmed RSV LRTD, Season 3 (Annual revaccination) |  | 37 |  | 6
Statistical Analysis 1: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD over season 1 in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 80.64, 95% CI 2-sided [55.90 to 92.73] — VE is defined as 1 minus the relative risk (RR). RR=the ratio of the incidence rates of RSVPreF3 Group over Placebo Group. VE (% ) = Vaccine Efficacy (Poisson method - adjusted by age, and region)
Statistical Analysis 2: Comparison: Placebo Group vs RSV_1_dose Group; To evaluate the efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD over season 2 in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 61.39, 95% CI 2-sided [36.44 to 77.70] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Placebo Group vs RSV_1_dose Group; To evaluate the efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD over season 3 in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 47.15, 95% CI 2-sided [7.06 to 71.59] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Placebo Group vs RSV_annual Group; To evaluate the efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD over season 2 in adults ≥ 60 YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 54.92, 95% CI 2-sided [27.85 to 72.98] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 5: Comparison: Placebo Group vs RSV_annual Group; To evaluate the efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD over season 3 in adults ≥ 60 YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 67.51, 95% CI 2-sided [22.35 to 88.79] — [estimate comment as in outcome 8, analysis 1]

9. Secondary Outcome: Number of Participants With First Episode of RT-PCR Confirmed RSV A and/or B Associated LRTD by Year Following a Single Dose of the RSVPreF3 OA Vaccine and Following Annual Revaccination Doses
Description: Efficacy of a single dose of the RSVPreF3 OA vaccine and annual revaccination doses was assessed against RSV A and/or B confirmed LRTD episode according to the case definition, by years after vaccination as follows: VE at each year includes the first occurrence of episodes reported from Day 14 post vaccination at first year, and for the next years, excluding analysis of participants who already reported a case in the previous year.
Time Frame: From Day 15 post first dose and each revaccination dose up to next dose or end of study (assessed approximately over a year after each vaccination [at Year 1, Year 2 and Year 3])
Population: Analysis was performed on the mES-RSV. Only participants with data available at specified timepoints were included in analysis. Analysis is presented based on the groups at each season (RSVPreF3 group for Year 1, RSV_1_dose and RSV_annual groups for Years 2 and 3, Placebo group for Years 1, 2 and 3).
Measure: Count of Participants; unit: Participants
Groups:
- RSV_1_dose Group: Participants received a dose of placebo every subsequent year.
- RSV_annual Group: Participants received an additional dose of RSVPreF3 OA vaccine every subsequent year
Arm/Group | RSVPreF3 Group | Placebo Group | RSV_1_dose Group | RSV_annual Group
Number analyzed (Participants) | 12468 | 12498 | 4988 | 4968
Participants
  RT-PCR-confirmed RSV LRTD, Year 1: number analyzed (Participants) | 12468 | 12498 | 0 | 0
  RT-PCR-confirmed RSV LRTD, Year 1 | 10 | 47 |  |
  RT-PCR-confirmed RSV LRTD, Year 2 (Single dose): number analyzed (Participants) | 0 | 10031 | 4988 | 0
  RT-PCR-confirmed RSV LRTD, Year 2 (Single dose) |  | 106 | 22 |
  RT-PCR-confirmed RSV LRTD, Year 2 (Annual revaccination): number analyzed (Participants) | 0 | 10031 | 0 | 4968
  RT-PCR-confirmed RSV LRTD, Year 2 (Annual revaccination) |  | 106 |  | 22
  RT-PCR-confirmed RSV LRTD, Year 3 (Single dose): number analyzed (Participants) | 0 | 10031 | 4988 | 0
  RT-PCR-confirmed RSV LRTD, Year 3 (Single dose) |  | 61 | 16 |
  RT-PCR-confirmed RSV LRTD, Year 3 (Annual revaccination): number analyzed (Participants) | 0 | 7224 | 0 | 3582
  RT-PCR-confirmed RSV LRTD, Year 3 (Annual revaccination) |  | 38 |  | 6
Statistical Analysis 1: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD over Year 1 in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 78.86, 95% CI 2-sided [57.62 to 90.48] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Placebo Group vs RSV_1_dose Group; To evaluate the efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD over Year 2 in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 58.59, 95% CI 2-sided [34.00 to 75.10] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Placebo Group vs RSV_1_dose Group; To evaluate the efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD over Year 3 in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 47.91, 95% CI 2-sided [8.51 to 71.97] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Placebo Group vs RSV_annual Group; To evaluate the efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD over Year 2 in adults ≥ 60 YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 58.33, 95% CI 2-sided [33.59 to 74.94] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 5: Comparison: Placebo Group vs RSV_annual Group; To evaluate the efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD over Year 3 in adults ≥ 60 YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 68.40, 95% CI 2-sided [24.64 to 89.08] — [estimate comment as in outcome 8, analysis 1]

10. Secondary Outcome: Number of Participants With First Episode of RT-PCR Confirmed RSV A and /or B Associated LRTD, Following a Single Dose of the RSVPreF3 OA Vaccine and Following Annual Revaccination Doses
Time Frame: From Day 15 post first dose to the first occurrence of RSV LRTD (assessed approximately over 3 years in the NH and 2.5-3 years in SH)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 12468 | 12498
Participants
  Season 1 | 10 | 47
  Season 2 (Single dose) | 32 | 154
  Season 2 (Annual revaccination) | 32 | 154
  Season 3 (NH) (Single dose) | 48 | 215
  Season 3 (NH) (Annual revaccination) | 38 | 192
Statistical Analysis 1: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the evolution of efficacy of a single dose of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD in adults ≥ 60 YOA over Season 1; Test type: Other — [test comment as in outcome 6, analysis 1]; Regression, Cox; VE = 78.75, 95% CI 2-sided [57.95 to 89.26] — VE is defined as 1 minus the relative risk (RR). RR=the ratio of the incidence rates of RSVPreF3 Group over Placebo Group. VE (%) = Vaccine Efficacy (Piecewise Cox model with time-varying efficacy - adjusted by age and region)
Statistical Analysis 2: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the evolution of efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD in adults ≥ 60 YOA over Season 2, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Regression, Cox; VE = 67.63, 95% CI 2-sided [52.47 to 77.95] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the evolution of efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD in adults ≥ 60 YOA over Season 3, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Regression, Cox; VE = 62.87, 95% CI 2-sided [46.76 to 74.11] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the evolution of efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD in adults ≥ 60 YOA over Season 2, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Regression, Cox; VE = 67.49, 95% CI 2-sided [52.27 to 77.86] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 5: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the evolution of efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD in adults ≥ 60 YOA over Season 3, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Regression, Cox; VE = 67.66, 95% CI 2-sided [51.71 to 78.34] — [estimate comment as in outcome 10, analysis 1]

11. Secondary Outcome: Number of Participants With First Episode of RT-PCR Confirmed RSV A and/or B Associated LRTD by Baseline Comorbidities Using Charlson Comorbidity Index Following a Single Dose of the RSVPreF3 OA Vaccine and Following Annual Revaccination Doses
Description: Efficacy of a single dose of the RSVPreF3 OA vaccine and annual revaccination doses is assessed against RSV A and/or B associated LRTD episode by baseline comorbidities using Charlson Comorbidity Index. Low/medium Risk = Participants with co-morbidity score at baseline less than or equal to 3 (Charlson Index); High Risk = Participants with co-morbidity score at baseline greater than 3 (Charlson Index).
Time Frame: as for outcome 7
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 8126 | 8268
Participants
  RT-PCR-confirmed RSV LRTD (Single dose), Low/Medium risk | 24 | 119
  RT-PCR-confirmed RSV LRTD (Single dose), High risk: number analyzed (Participants) | 4342 | 4230
  RT-PCR-confirmed RSV LRTD (Single dose), High risk | 24 | 96
  RT-PCR-confirmed RSV LRTD (Annual revaccination), Low/Medium risk | 18 | 108
  RT-PCR-confirmed RSV LRTD (Annual revaccination), High risk: number analyzed (Participants) | 4342 | 4230
  RT-PCR-confirmed RSV LRTD (Annual revaccination), High risk | 20 | 84
Statistical Analysis 1: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD in adults ≥ 60 YOA by baseline comorbidities with low/medium risk (Charlson Comorbidity Index), following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 66.49, 95% CI 2-sided [47.54 to 79.40] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD in adults ≥ 60 YOA by baseline comorbidities with high risk (Charlson Comorbidity Index), following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 58.88, 95% CI 2-sided [34.81 to 74.98] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD in adults ≥ 60 YOA by baseline comorbidities with low/medium risk (Charlson Comorbidity Index), following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 72.55, 95% CI 2-sided [54.34 to 84.37] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD in adults ≥ 60 YOA by baseline comorbidities with high risk (Charlson Comorbidity Index), following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 61.99, 95% CI 2-sided [37.17 to 78.01] — [estimate comment as in outcome 4, analysis 1]

12. Secondary Outcome: Number of Participants With First Episode of RT-PCR Confirmed RSV A and/or B Associated LRTD by Baseline Comorbidities According to Comorbidities of Interest Following a Single Dose of the RSVPreF3 OA Vaccine and Following Annual Revaccination Doses
Description: Efficacy of a single dose of the RSVPreF3 OA vaccine and annual revaccination doses is assessed against RSV A and/or B associated LRTD episode by baseline comorbidities of interest divided into 2: cardiorespiratory conditions such as chronic obstructive pulmonary disease (COPD), asthma, any chronic respiratory or pulmonary disease, and endocrinometabolic conditions such as diabetes mellitus type 1 or 2, chronic heart failure and advanced liver or renal disease.
Time Frame: as for outcome 7
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 7454 | 7547
Participants
  Confirmed RSV LRTD (Single dose), No pre-existing comorbidity of interest | 23 | 99
  Confirmed RSV LRTD (Single dose), At least 1 pre-existing comorbidity of interest: number analyzed (Participants) | 5014 | 4951
  Confirmed RSV LRTD (Single dose), At least 1 pre-existing comorbidity of interest | 25 | 116
  Confirmed RSV LRTD (Single dose), At least 1 pre-existing Cardiorespiratory condition: number analyzed (Participants) | 2577 | 2504
  Confirmed RSV LRTD (Single dose), At least 1 pre-existing Cardiorespiratory condition | 17 | 85
  Confirmed RSV LRTD (Single dose), At least 1 pre-existing Endocrinometabolic condition: number analyzed (Participants) | 3243 | 3274
  Confirmed RSV LRTD (Single dose), At least 1 pre-existing Endocrinometabolic condition | 12 | 55
  Confirmed RSV LRTD (Annual revaccination), No pre-existing comorbidity of interest | 20 | 91
  Confirmed RSV LRTD (Annual revaccination), At least 1 pre-existing comorbidity of interest: number analyzed (Participants) | 5014 | 4951
  Confirmed RSV LRTD (Annual revaccination), At least 1 pre-existing comorbidity of interest | 18 | 101
  Confirmed RSV LRTD (Annual revaccination), At least 1 pre-existing Cardiorespiratory condition: number analyzed (Participants) | 2577 | 2504
  Confirmed RSV LRTD (Annual revaccination), At least 1 pre-existing Cardiorespiratory condition | 11 | 73
  Confirmed RSV LRTD (Annual revaccination), At least 1 pre-existing Endocrinometabolic condition: number analyzed (Participants) | 3243 | 3274
  Confirmed RSV LRTD (Annual revaccination), At least 1 pre-existing Endocrinometabolic condition | 9 | 49
Statistical Analysis 1: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD in adults ≥ 60 YOA with no pre-existing comorbidity of interest, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 61.48, 95% CI 2-sided [38.62 to 76.74] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD in adults ≥ 60 YOA with at least 1 pre-existing comorbidity of interest, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 64.73, 95% CI 2-sided [45.10 to 78.14] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD in adults ≥ 60 YOA with at least 1 pre-existing cardiorespiratory condition, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 68.14, 95% CI 2-sided [45.71 to 82.33] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD in adults ≥ 60 YOA with at least 1 pre-existing endocrinometabolic condition, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 63.88, 95% CI 2-sided [31.35 to 82.48] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD in adults ≥ 60 YOA with no pre-existing comorbidity of interest, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 64.16, 95% CI 2-sided [41.08 to 79.17] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD in adults ≥ 60 YOA with at least 1 pre-existing comorbidity of interest, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 71.19, 95% CI 2-sided [51.92 to 83.65] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD in adults ≥ 60 YOA with at least 1 pre-existing cardiorespiratory condition,following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 75.94, 95% CI 2-sided [54.11 to 88.54] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD in adults ≥ 60 YOA with at least 1 pre-existing endocrinometabolic condition, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 69.85, 95% CI 2-sided [37.51 to 87.05] — [estimate comment as in outcome 4, analysis 1]

13. Secondary Outcome: Number of Participants With First Episode of RT-PCR Confirmed RSV A and/or B Associated LRTD by Baseline Frailty Status Following a Single Dose of the RSVPreF3 OA Vaccine and Following Annual Revaccination Doses
Description: Efficacy of a single dose of the RSVPreF3 OA vaccine and annual revaccination doses is assessed against RSV A and /or B associated LRTD episode according to the case definition, by baseline frailty status of frail, pre-frail and fit. Frail = Participants with a walking speed of less than (<) 0.4 meters per second (m/s) or who were not able to perform the test; Pre-Frail = Participants with a walking speed between 0.4-0.99 m/s; Fit = Participants with a walking speed of ≥1 m/s.
Time Frame: as for outcome 7
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 7464 | 7523
Participants
  RT-PCR-confirmed RSV LRTD (Single dose), Frail: number analyzed (Participants) | 189 | 176
  RT-PCR-confirmed RSV LRTD (Single dose), Frail | 2 | 1
  RT-PCR-confirmed RSV LRTD (Single dose), Pre-Frail: number analyzed (Participants) | 4794 | 4779
  RT-PCR-confirmed RSV LRTD (Single dose), Pre-Frail | 12 | 67
  RT-PCR-confirmed RSV LRTD (Single dose), Fit | 34 | 145
  RT-PCR-confirmed RSV LRTD (Annual revaccination), Frail: number analyzed (Participants) | 189 | 176
  RT-PCR-confirmed RSV LRTD (Annual revaccination), Frail | 1 | 1
  RT-PCR-confirmed RSV LRTD (Annual revaccination), Pre-Frail: number analyzed (Participants) | 4794 | 4779
  RT-PCR-confirmed RSV LRTD (Annual revaccination), Pre-Frail | 10 | 63
  RT-PCR-confirmed RSV LRTD (Annual revaccination), Fit | 27 | 126
Statistical Analysis 1: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD by baseline frailty status (frail) in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = -153.57, 95% CI 2-sided [-16322.97 to 88.00] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD by baseline frailty status (pre-frail) in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 70.07, 95% CI 2-sided [43.89 to 85.33] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD by baseline frailty status (fit) in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 61.04, 95% CI 2-sided [42.89 to 74.08] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD by baseline frailty status (frail) in adults ≥ 60 YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 13.62, 95% CI 2-sided [-6751.38 to 98.91] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD by baseline frailty status (pre-frail) in adults ≥ 60 YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 74.32, 95% CI 2-sided [49.33 to 88.31] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed LRTD by baseline frailty status (fit) in adults ≥ 60 YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 64.79, 95% CI 2-sided [46.10 to 77.75] — [estimate comment as in outcome 4, analysis 1]

14. Secondary Outcome: Number of Participants With First Episode of RT-PCR Confirmed RSV A and/or B Associated Severe LRTD Following a Single Dose of the RSVPreF3 OA Vaccine and Following Annual Revaccination Doses
Description: Efficacy of a single dose of the RSVPreF3 OA vaccine and annual revaccination doses is assessed against RSV A and/or B associated severe LRTD episode. Case definition for RSV-confirmed severe LRTD: An RT-PCR confirmed case of RSV-associated severe LRTD is characterized by presence of lower respiratory signs or an LRTD episode assessed as severe by the investigator (Severe LRTD case definition 1) or presence of an LRTD with need for oxygen supplementation or need for positive airway pressure therapy or need for other types of mechanical ventilation (Severe LRTD case definition 2) and with at least one RSV positive swab detected by RT-PCR.
Time Frame: as for outcome 7
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 12468 | 12498
Participants
  RT-PCR-confirmed RSV severe LRTD (Single dose), Any | 15 | 75
  RT-PCR-confirmed RSV severe LRTD (Single dose), Definition 1: Clinical symptomology | 15 | 75
  RT-PCR-confirmed RSV severe LRTD (Single dose), Definition 2: Supportive therapy | 2 | 7
  RT-PCR-confirmed RSV severe LRTD (Annual revaccination), Any | 9 | 67
  RT-PCR-confirmed RSV severe LRTD (Annual revaccination), Definition 1: Clinical symptomology | 9 | 67
  RT-PCR-confirmed RSV severe LRTD (Annual revaccination), Definition 2: Supportive therapy | 0 | 6
Statistical Analysis 1: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of severe RSV-confirmed LRTD in adults ≥ 60 YOA according to any case definition, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 67.38, 95% CI 2-sided [42.43 to 82.68] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of severe RSV-confirmed LRTD in adults ≥ 60 YOA according to case definition 1, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 67.38, 95% CI 2-sided [42.43 to 82.68] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of severe RSV-confirmed LRTD in adults ≥ 60 YOA according to the case definition 2, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 59.16, 95% CI 2-sided [-119.60 to 95.93] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of severe RSV-confirmed LRTD in adults ≥ 60 YOA according to any case definition, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 78.80, 95% CI 2-sided [57.05 to 90.75] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of severe RSV-confirmed LRTD in adults ≥ 60 YOA according to case definition 1, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 78.80, 95% CI 2-sided [57.05 to 90.75] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of severe RSV-confirmed LRTD in adults ≥ 60 YOA according to case definition 2, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 100.00, 95% CI 2-sided [20.27 to 100.00] — [estimate comment as in outcome 4, analysis 1]

15. Secondary Outcome: Number of Participants With First Episode of RT-PCR Confirmed RSV A and/or B Associated ARI Following a Single Dose of the RSVPreF3 OA Vaccine and Following Annual Revaccination Doses
Description: Efficacy of a single dose of the RSVPreF3 OA vaccine and annual revaccination doses is assessed against RSV confirmed A and/or B associated ARI episode. A case of RT-PCR confirmed RSV-associated ARI is characterized by the presence of respiratory symptoms/signs for at least 24 hours OR respiratory symptom/sign + systemic symptom/sign for at least 24 hours with at least one RSV-positive swab detected by RT-PCR.
Time Frame: as for outcome 7
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 12468 | 12498
Participants
  RT-PCR-confirmed RSV ARI (Single dose) | 131 | 428
  RT-PCR-confirmed RSV ARI (Annual revaccination) | 103 | 385
Statistical Analysis 1: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed ARI in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 51.13, 95% CI 2-sided [40.31 to 60.21] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of RSV-confirmed ARI in adults ≥ 60 YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 58.44, 95% CI 2-sided [48.10 to 66.96] — [estimate comment as in outcome 4, analysis 1]

16. Secondary Outcome: Number of Participants With First Episode of Any ARI or Any LRTD Following a Single Dose of the RSVPreF3 OA Vaccine and Following Annual Revaccination Doses
Description: Efficacy of a single dose of the RSVPreF3 OA vaccine and annual revaccination doses is assessed against any ARI and any LRTD.
Time Frame: From Day 15 post first vaccination up to study end (approximately 3 years for NH and 2.5-3 years for SH)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 12469 | 12503
Participants
  Any ARI (Single dose) | 4858 | 6096
  Any ARI (Annual revaccination) | 4731 | 5914
  Any LRTD (Single dose) | 12450 | 3352
  Any LRTD (Annual revaccination) | 2308 | 3210
Statistical Analysis 1: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of any ARI in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 2.33, 95% CI 2-sided [-1.47 to 5.99] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of any ARI in adults ≥ 60 YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 3.32, 95% CI 2-sided [-0.50 to 6.98] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of any LRTD in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 3.68, 95% CI 2-sided [-1.55 to 8.63] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of any LRTD in adults ≥ 60 YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 6.99, 95% CI 2-sided [1.81 to 11.90] — [estimate comment as in outcome 4, analysis 1]

17. Secondary Outcome: Number of Hospitalizations Due to RSV-confirmed Respiratory Diseases or Due to Complication Related to RSV-confirmed Respiratory Diseases, Following a Single Dose of the RSVPreF3 OA Vaccine and Following Annual Revaccination Doses up to End of Study
Description: RSV infection was confirmed by RT-PCR.
Time Frame: From Day 15 post-first vaccination up to study end (approximately 3 years for NH and 2.5-3 years for SH)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 12468 | 12498
Participants
  RSV respiratory disease (Single dose), during season | 2 | 4
  RSV respiratory disease or related complication (Single dose), during season | 2 | 4
  RSV respiratory disease (Annual revaccination),during season | 0 | 4
  RSV respiratory disease or related complication (Annual revaccination), during season | 0 | 4
  RSV respiratory disease (Single dose), up to end of study | 2 | 6
  RSV respiratory disease or related complication (Single dose), up to end of study | 2 | 6
  RSV respiratory disease (Annual revaccination), up to end of study | 0 | 6
  RSV respiratory disease or related complication (Annual revaccination), up to end of study | 0 | 6
Statistical Analysis 1: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of hospitalization due to RT-PCR-confirmed RSV respiratory disease during the study period in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 50.37, 95% CI 2-sided [-184.45 to 95.19] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of hospitalization due to RT-PCR-confirmed RSV respiratory disease or complication related to RT-PCR-confirmed RSV ARI during the study period in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 50.37, 95% CI 2-sided [-184.45 to 95.19] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of hospitalization due to RT-PCR-confirmed RSV respiratory disease during the study period in adults ≥ 60 YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 100.00, 95% CI 2-sided [11.56 to 100.00] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of hospitalization due to RT-PCR-confirmed RSV respiratory disease or complication related to RT-PCR-confirmed RSV ARI during the study period in adults ≥ 60 YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 100.00, 95% CI 2-sided [11.56 to 100.00] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of hospitalization due to RT-PCR-confirmed RSV respiratory disease during the RSV seson in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 22.14, 95% CI 2-sided [-457.67 to 93.12] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of hospitalization due to RT-PCR-confirmed RSV respiratory disease or complication related to RT-PCR-confirmed RSV ARI during the RSV season in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 22.14, 95% CI 2-sided [-457.67 to 93.12] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of hospitalization due to RT-PCR-confirmed RSV respiratory disease during the RSV season in adults ≥ 60 YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 100.00, 95% CI 2-sided [-54.53 to 100.00] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of hospitalization due to RT-PCR-confirmed RSV respiratory disease or complication related to RT-PCR-confirmed RSV ARI during the RSV season in adults ≥ 60 YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 100.00, 95% CI 2-sided [-54.53 to 100.00] — [estimate comment as in outcome 4, analysis 1]

18. Secondary Outcome: Number of Hospitalizations Due to Any Respiratory Diseases or Due to a Complication Related to Any Respiratory Diseases, During the RSV Seasons Following a Single Dose of the RSVPreF3 OA Vaccine and Following Annual Revaccination Doses up to End of Study
Description: A diagnosis of respiratory disease included: acute respiratory infections, other diseases of upper respiratory tract, pneumonia and influenza, chronic obstructive pulmonary disease and allied conditions, pneumoconioses and other lung diseases due to external agents, other diseases of respiratory system.
Time Frame: From Day 15 post-first vaccination up to study end (approximately 3 years for NH and 2.5-3 years for SH)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 12469 | 12503
Participants
  Any respiratory disease (Single dose), during seasons: number analyzed (Participants) | 12468 | 12498
  Any respiratory disease (Single dose), during seasons | 121 | 174
  Any respiratory disease or related complication (Single dose), during seasons: number analyzed (Participants) | 12468 | 12498
  Any respiratory disease or related complication (Single dose), during seasons | 131 | 180
  Any respiratory disease (Annual revaccination), during seasons: number analyzed (Participants) | 12468 | 12498
  Any respiratory disease (Annual revaccination), during seasons | 114 | 163
  Any respiratory disease or related complication (Annual revaccination), during seasons: number analyzed (Participants) | 12468 | 12498
  Any respiratory disease or related complication (Annual revaccination), during seasons | 119 | 169
  Any respiratory disease (Single dose), up to end of study | 167 | 221
  Any respiratory disease or related complication (Single dose), up to end of study | 179 | 230
  Any respiratory disease (Annual revaccination), up to end of study | 163 | 208
  Any respiratory disease or related complication (Annual revaccination), up to end of study | 171 | 217
Statistical Analysis 1: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of hospitalization due to any respiratory diseases during the study period in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = -1.81, 95% CI 2-sided [-25.43 to 17.49] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of hospitalization due to any respiratory diseases or complication related to any respiratory disease during the study period in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = -4.72, 95% CI 2-sided [-28.26 to 14.61] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of hospitalization due to any respiratory diseases during the study period in adults ≥ 60 YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = -3.61, 95% CI 2-sided [-28.20 to 16.38] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of hospitalization due to any respiratory diseases or complication related to any respiratory diseases during the study period in adults ≥ 60 YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = -3.59, 95% CI 2-sided [-27.55 to 15.98] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of hospitalization due to any respiratory diseases during the RSV season in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 2.98, 95% CI 2-sided [-23.52 to 23.99] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of hospitalization due to any respiratory diseases or complication related to any respiratory disease during the RSV seasons in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = -1.71, 95% CI 2-sided [-28.56 to 19.70] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of hospitalization due to any respiratory diseases during the RSV seasons in adults ≥ 60 YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 4.80, 95% CI 2-sided [-22.14 to 26.00] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of hospitalization due to any respiratory diseases or complication related to any respiratory diseases during the RSV seasons in adults ≥ 60 YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 4.64, 95% CI 2-sided [-21.73 to 25.48] — [estimate comment as in outcome 4, analysis 1]

19. Secondary Outcome: Number of Complications Related to RSV-confirmed ARI During the RSV Seasons Following a Single Dose of the RSVPreF3 OA Vaccine and Following Annual Revaccination Doses up to End of Study
Description: RSV infection was confirmed by RT-PCR.
Time Frame: From Day 15 post-first vaccination up to study end (approximately 3 years for NH and 2.5-3 years for SH)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 12468 | 12498
Participants
  Related to RT-PCR-confirmed RSV ARI (Single dose), up to end of study | 12 | 50
  Related to RT-PCR-confirmed RSV ARI (Annual revaccination), up to end of study | 11 | 46
  Related to RT-PCR-confirmed RSV ARI (Single dose), during season | 9 | 43
  Related to RT-PCR-confirmed RSV ARI (Annual revaccination), during season | 9 | 39
Statistical Analysis 1: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of complications related to RSV- ARI during the study period in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 62.94, 95% CI 2-sided [28.91 to 82.15] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of complications related to RSV-ARI during the study period in adults ≥ 60 YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 63.80, 95% CI 2-sided [28.50 to 83.20] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of complications related to RSV- ARI during the RSV seasons in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 65.69, 95% CI 2-sided [28.56 to 85.47] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of complications related to RSV-ARI during the RSV seasons in adults ≥ 60 YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 62.87, 95% CI 2-sided [21.45 to 84.29] — [estimate comment as in outcome 4, analysis 1]

20. Secondary Outcome: Number of Complications Related to Any ARI During the RSV Seasons Following a Single Dose of the RSVPreF3 OA Vaccine and Following Annual Revaccination Doses up to End of Study
Description: RSV infection was confirmed by RT-PCR.
Time Frame: From Day 15 post-first vaccination up to study end (approximately 3 years for NH and 2.5-3 years for SH)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 12469 | 12503
Participants
  Complications related to any ARI (Single dose), during season | 438 | 695
  Complications related to any ARI (Annual revaccination), during season | 417 | 660
  Complications related to any ARI (Single dose), up to end of study | 620 | 863
  Complications related to any ARI (Annual revaccination), up to end of study | 579 | 823
Statistical Analysis 1: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of complications related to any ARI during the study period in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 2.59, 95% CI 2-sided [-8.29 to 12.42] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of complications related to any ARI during the study period in adults ≥ 60 YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 6.70, 95% CI 2-sided [-4.05 to 16.39] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of complications related to any ARI during the RSV seasons in adults ≥ 60 YOA, following a single dose of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 10.95, 95% CI 2-sided [-0.68 to 21.31] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: RSVPreF3 Group vs Placebo Group; To evaluate the vaccine efficacy of the RSVPreF3 OA investigational vaccine in the prevention of complications related to any ARI during the RSV seasons in adults ≥ 60 YOA, following annual revaccination of the RSVPreF3 OA investigational vaccine; Test type: Other — [test comment as in outcome 6, analysis 1]; Poisson regression method; VE = 12.12, 95% CI 2-sided [0.32 to 22.58] — [estimate comment as in outcome 4, analysis 1]

21. Secondary Outcome: Maximum Influenza Patient-Reported Outcome (Flu-PRO) Chest Score for the Participants With RT-PCR-confirmed RSV A and/or B-associated ARI Following a Single Dose of the RSVPreF3 OA Vaccine and Following Annual Revaccination Doses
Description: For this outcome measure, the Health Related -Quality of life (HR-QOL) score is measured by Flu-PRO questionnaire version 2.0. The Flu-PRO is a 32 items daily diary, which assesses influenza signs across 6 body systems- nose, throat, eyes, chest/respiratory, gastrointestinal and body/systemic. The objective of this outcome measure was to present data only for chest/respiratory system after a single dose and after annual revaccination. The FLU-PRO score was computed as the mean score across questionaire items for chest/respiratory body system, with the scores ranging from 0 (symptom free) to 4 (very severe symptoms).
Time Frame: During the first 7 days from the onset of ARI symptoms (assessed from Day 15 post first vaccination dose until end of study [approximately 3 years in NH and 2.5-3 years in SH])
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 121 | 377
Scores on a scale
  Chest / Respiratory (Single dose) | 1.60 (0.89) | 1.97 (0.88)
  Chest / Respiratory (Annual revaccination): number analyzed (Participants) | 97 | 341
  Chest / Respiratory (Annual revaccination) | 1.50 (0.87) | 1.96 (0.89)

22. Secondary Outcome: Least Square Mean Flu-PRO Total Score for the Participants With RT-PCR-confirmed RSV A and/or B-associated ARI Following a Single Dose of the RSVPreF3 OA Vaccine and Following Annual Revaccination Doses
Description: The Flu-PRO questionnaire version 2.0 is a 32 items daily diary, which assesses influenza signs across 6 body systems- nose, throat, eyes, chest/respiratory, gastrointestinal and body/systemic. The FLU-PRO total score was computed as the mean score across all 32 items of the questionaire for all 6 body systems, with the total scores ranging from 0 (symptom free) to 4 (very severe symptoms).
Time Frame: as for outcome 21
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 131 | 428
Scores on a scale
  Day 1 to Day 7 (Single dose) | 0.85 (0.07) | 0.92 (0.06)
  Day 1 to Day 7 (Annual revaccination): number analyzed (Participants) | 103 | 385
  Day 1 to Day 7 (Annual revaccination) | 0.81 (0.07) | 0.90 (0.06)

23. Secondary Outcome: EuroQol 5-dimension Health Questionnaire (EQ-5D) Utility Score for Participants With RT-PCR-confirmed RSV A and/or B-associated ARI Following a Single Dose of the RSVPreF3 OA Vaccine and Following Annual Revaccination Doses
Description: The EQ-5D is a general health utility questionnaire with health states, defined through 5 dimensions- mobility, self-care, usual activities, pain/ discomfort and anxiety/ depression. A participant who responds 1 (no problem/no symptom) to all 5 items has a profile "11111" and similarly a participant who responds 3 (the highest level of difficulty or symptom) to all items has a profile "33333". The health states indicated in these 5 dimensions are converted and presented as a single mean index value as recommended by EuroQol group, where values range from 0 (worst) to 1 (full health).
Time Frame: At the ARI visit (assessed from Day 15 post first vaccination dose until end of study- approximately 3 years in NH and 2.5-3 years in SH)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 106 | 362
Scores on a scale
  At ARI visit (Single dose) | 0.8164 (0.0258) | 0.7886 (0.0197)
  At ARI visit (Annual revaccination): number analyzed (Participants) | 85 | 324
  At ARI visit (Annual revaccination) | 0.8377 (0.0259) | 0.7966 (0.0197)

24. Secondary Outcome: Least Square Mean of Short Form-12 (SF-12) Health Survey for Participants With RT-PCR Confirmed RSV A and/or B-associated ARI Following a Single Dose of the RSVPreF3 OA Vaccine and Following Annual Revaccination Doses
Description: SF-12 is a health survey with 12 questions, covering 8 domains- physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health. Summary scores are computed from these domains for the physical and mental component. The total score of the SF-12 questionnaire is evaluated on a scale from 0 to 100, with a higher score indicating a better perceived health-related quality of life.
Time Frame: At the ARI visit (assessed from one-month post first vaccination dose until end of study- approximately 3 years in NH and 2.5-3 years in SH)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 105 | 361
Scores on a scale
  At ARI visit (Single dose) | 59.43 (4.07) | 57.51 (3.15)
  At ARI visit (Annual revaccination): number analyzed (Participants) | 88 | 322
  At ARI visit (Annual revaccination) | 63.65 (4.15) | 59.02 (3.18)

25. Secondary Outcome: Duration in Days of RT-PCR Confirmed RSV A and/or B ARI and LRTD Episodes
Description: The duration in days of RT-PCR confirmed RSV A and/or B ARI and LRTD episodes are described.
Time Frame: From Day 15 post first dose to end of Season 1, from 15 days post-second dose administration to end of Season 2, and from start to end of Season 3 [all seasons summing approximately 3 years in NH and 2.5-3 years in SH]
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | RSVPreF3 Group | Placebo Group | RSV_1_dose Group | RSV_annual Group
Number analyzed (Participants) | 40 | 208 | 61 | 45
Days
  RT-PCR-confirmed RSV ARI, Season 1: number analyzed (Participants) | 40 | 111 | 0 | 0
  RT-PCR-confirmed RSV ARI, Season 1 | 12.0 [8.0 to 19.0] | 15.0 [11.0 to 22.0] |  |
  RT-PCR-confirmed RSV LRTD, Season 1: number analyzed (Participants) | 10 | 47 | 0 | 0
  RT-PCR-confirmed RSV LRTD, Season 1 | 15.5 [8.0 to 19.0] | 20.0 [15.0 to 27.0] |  |
  RT-PCR-confirmed RSV ARI, Season 2: number analyzed (Participants) | 0 | 208 | 61 | 45
  RT-PCR-confirmed RSV ARI, Season 2 |  | 16.0 [12.0 to 24.0] | 14.0 [10.0 to 23.0] | 13.0 [9.0 to 18.0]
  RT-PCR-confirmed RSV LRTD, Season 2: number analyzed (Participants) | 0 | 107 | 22 | 22
  RT-PCR-confirmed RSV LRTD, Season 2 |  | 16.0 [13.0 to 24.0] | 17.0 [10.0 to 28.0] | 14.0 [9.0 to 23.0]
  RT-PCR-confirmed RSV ARI, Season 3: number analyzed (Participants) | 0 | 111 | 29 | 19
  RT-PCR-confirmed RSV ARI, Season 3 |  | 16.0 [14.0 to 22.0] | 16.0 [13.0 to 24.0] | 10.0 [7.0 to 21.0]
  RT-PCR-confirmed RSV LRTD, Season 3: number analyzed (Participants) | 0 | 60 | 16 | 6
  RT-PCR-confirmed RSV LRTD, Season 3 |  | 17.5 [14.5 to 26.0] | 16.5 [15.0 to 24.5] | 12.0 [7.0 to 21.0]

26. Secondary Outcome: Number of Participants With Each Reported Symptom/Sign and Supportive Therapy Use Associated With of RT-PCR Confirmed RSV A and/or B ARI Episodes During Season 1
Description: RSV infection was confirmed by RT-PCR, and the symptoms/signs and supportive therapy use associated with RT-PCR confirmed RSV A and/or RSV B ARI episodes were reported. Fever was defined as a temperature ≥38.0 degrees Celsius (°C) by any route.
Time Frame: From Day 15 post-dose 1 administration up to end of season 1 in the SH [a median of approximately 11.5 months (11.6 months in NH and 9.1 months in SH)]
Population: Analysis was performed on the mES. Only participants with data available for symptoms/signs and supportive therapy use associated with RT-PCR confirmed RSV A and/or RSV B ARI episodes at specified timepoints were included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 40 | 110
Participants
  Nasal Congestion | 28 | 83
  Rhinorrhea: number analyzed (Participants) | 39 | 110
  Rhinorrhea | 32 | 93
  Sore Throat | 26 | 76
  Cough (new or increased) | 36 | 101
  Sputum (new or increased) | 20 | 75
  Shortness of breath or dyspnea (new or increased) | 7 | 35
  Wheezing (new or increased): number analyzed (Participants) | 40 | 109
  Wheezing (new or increased) | 5 | 25
  Crackles: number analyzed (Participants) | 38 | 105
  Crackles | 1 | 6
  Rhonchi: number analyzed (Participants) | 38 | 105
  Rhonchi | 1 | 13
  Respiratory rate ≥20 breaths/minute: number analyzed (Participants) | 39 | 106
  Respiratory rate ≥20 breaths/minute | 3 | 11
  Low or decreased oxygen saturation: number analyzed (Participants) | 39 | 105
  Low or decreased oxygen saturation | 1 | 9
  Fever: number analyzed (Participants) | 40 | 107
  Fever | 2 | 8
  Feverishness | 8 | 24
  Fatigue | 22 | 67
  Body aches | 12 | 40
  Headache | 20 | 55
  Decreased appetite | 13 | 42
  Need for oxygen supplementation | 0 | 4
  Need for positive airway pressure therapy | 0 | 0
  Need of other types of mechanical ventilation | 0 | 0
  Other symptoms or signs | 7 | 22

27. Secondary Outcome: Number of Participants With Each Reported Symptom/Sign and Supportive Therapy Use Associated With of RT-PCR Confirmed RSV A and/or B ARI Episodes During Season 2
Description: as for outcome 26
Time Frame: From Day 15 post-dose 2 administration up to end of Season 2 in SH (a median of approximately 11.9 months [11.9 months in NH and 7.5 months in SH])
Population: Analysis was performed on the modified Exposed set for Dose 2 (mES-Dose 2), which included all participants who received the first and second doses of the study intervention, and who did not report an RSV-confirmed ARI prior to Day 15 after each vaccination. Only participants with data available for symptoms/signs and supportive therapy use associated with RT-PCR confirmed RSV A and/or RSV B ARI episodes at specified timepoints were included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | RSV_1_dose Group | RSV_annual Group
Number analyzed (Participants) | 208 | 61 | 45
Participants
  Nasal Congestion | 162 | 43 | 31
  Rhinorrhea | 186 | 52 | 39
  Sore Throat | 147 | 43 | 33
  Cough (new or increased) | 201 | 55 | 41
  Sputum (new or increased) | 150 | 39 | 29
  Shortness of breath or dyspnea (new or increased): number analyzed (Participants) | 207 | 61 | 45
  Shortness of breath or dyspnea (new or increased) | 79 | 17 | 19
  Wheezing (new or increased): number analyzed (Participants) | 207 | 61 | 45
  Wheezing (new or increased) | 56 | 15 | 10
  Crackles: number analyzed (Participants) | 197 | 60 | 44
  Crackles | 19 | 2 | 3
  Rhonchi: number analyzed (Participants) | 197 | 60 | 44
  Rhonchi | 32 | 8 | 7
  Respiratory rate ≥20 breaths/minute: number analyzed (Participants) | 201 | 61 | 45
  Respiratory rate ≥20 breaths/minute | 21 | 5 | 0
  Low or decreased oxygen saturation: number analyzed (Participants) | 201 | 61 | 45
  Low or decreased oxygen saturation | 8 | 1 | 4
  Fever: number analyzed (Participants) | 206 | 59 | 45
  Fever | 21 | 5 | 7
  Feverishness: number analyzed (Participants) | 208 | 60 | 45
  Feverishness | 64 | 13 | 15
  Fatigue | 145 | 34 | 33
  Body aches | 91 | 27 | 24
  Headache | 124 | 36 | 28
  Decreased appetite | 85 | 20 | 18
  Need for oxygen supplementation | 1 | 1 | 0
  Need for positive airway pressure therapy: number analyzed (Participants) | 207 | 60 | 45
  Need for positive airway pressure therapy | 0 | 1 | 0
  Need of other types of mechanical ventilation: number analyzed (Participants) | 208 | 60 | 45
  Need of other types of mechanical ventilation | 0 | 0 | 0
  Other symptoms or signs: number analyzed (Participants) | 207 | 61 | 45
  Other symptoms or signs | 48 | 12 | 14

28. Secondary Outcome: Number of Participants With Each Reported Symptom/Sign and Supportive Therapy Use Associated With of RT-PCR Confirmed RSV A and/or B ARI Episodes During Season 3
Description: as for outcome 26
Time Frame: From start of Season 3 up to end of Season 3 in NH (a median of approximately 7 months)
Population: Analysis was performed on the mES-Dose 2. Only participants with data available for symptoms/signs and supportive therapy use associated with RT-PCR confirmed RSV A and/or RSV B ARI episodes at specified timepoints were included in analysis. Only participants in NH were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | RSV_1_dose Group | RSV_annual Group
Number analyzed (Participants) | 113 | 30 | 19
Participants
  Nasal Congestion | 101 | 25 | 15
  Rhinorrhea | 98 | 26 | 17
  Sore Throat | 76 | 17 | 14
  Cough (new or increased) | 111 | 27 | 18
  Sputum (new or increased) | 86 | 23 | 10
  Shortness of breath or dyspnea (new or increased): number analyzed (Participants) | 111 | 30 | 19
  Shortness of breath or dyspnea (new or increased) | 42 | 10 | 5
  Wheezing (new or increased): number analyzed (Participants) | 112 | 30 | 19
  Wheezing (new or increased) | 32 | 6 | 3
  Crackles: number analyzed (Participants) | 111 | 27 | 19
  Crackles | 10 | 2 | 0
  Rhonchi: number analyzed (Participants) | 111 | 27 | 19
  Rhonchi | 16 | 8 | 2
  Respiratory rate ≥20 breaths/minute: number analyzed (Participants) | 112 | 27 | 19
  Respiratory rate ≥20 breaths/minute | 9 | 3 | 0
  Low or decreased oxygen saturation: number analyzed (Participants) | 112 | 27 | 19
  Low or decreased oxygen saturation | 11 | 1 | 3
  Fever | 10 | 2 | 0
  Feverishness | 32 | 14 | 6
  Fatigue | 85 | 21 | 15
  Body aches | 56 | 16 | 10
  Headache | 66 | 16 | 12
  Decreased appetite | 52 | 13 | 12
  Need for oxygen supplementation | 0 | 1 | 0
  Need for positive airway pressure therapy | 0 | 0 | 0
  Need of other types of mechanical ventilation | 0 | 0 | 0
  Other symptoms or signs | 35 | 6 | 9

29. Secondary Outcome: Number of Participants With Each Reported Symptom/Sign and Supportive Therapy Use Associated With of RT-PCR Confirmed RSV A and/or B LRTD Episodes During Season 1
Description: RSV infection was confirmed by RT-PCR, and the symptoms/signs and supportive therapy use associated with RT-PCR confirmed RSV A and/or RSV B LRTD episodes were reported. Fever was defined as a temperature ≥38.0°C by any route.
Time Frame: as for outcome 26
Population: Analysis was performed on the mES-RSV. Only participants with data available for symptoms/signs and supportive therapy use associated with RT-PCR confirmed RSV A and/or RSV B LRTD episodes at specified timepoints were included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 10 | 47
Participants
  Nasal Congestion | 7 | 38
  Rhinorrhea | 9 | 38
  Sore Throat | 5 | 33
  Cough (new or increased) | 10 | 47
  Sputum (new or increased) | 8 | 36
  Shortness of breath or dyspnea (new or increased) | 4 | 29
  Wheezing (new or increased) | 5 | 24
  Crackles: number analyzed (Participants) | 10 | 45
  Crackles | 1 | 6
  Rhonchi: number analyzed (Participants) | 10 | 45
  Rhonchi | 0 | 13
  Respiratory rate ≥20 breaths/minute: number analyzed (Participants) | 10 | 45
  Respiratory rate ≥20 breaths/minute | 3 | 10
  Low or decreased oxygen saturation: number analyzed (Participants) | 10 | 44
  Low or decreased oxygen saturation | 1 | 8
  Fever: number analyzed (Participants) | 10 | 46
  Fever | 1 | 8
  Feverishness | 2 | 16
  Fatigue | 6 | 37
  Body aches | 5 | 22
  Headache | 4 | 27
  Decreased appetite | 7 | 26
  Need for oxygen supplementation | 0 | 4
  Need for positive airway pressure therapy | 0 | 0
  Need of other types of mechanical ventilation | 0 | 0
  Other symptoms or signs | 2 | 12

30. Secondary Outcome: Number of Participants With Each Reported Symptom/Sign and Supportive Therapy Use Associated With of RT-PCR Confirmed RSV A and/or B LRTD Episodes During Season 2
Description: as for outcome 29
Time Frame: as for outcome 27
Population: Analysis was performed on the mES-Dose 2. Only participants with data available for symptoms/signs and supportive therapy use associated with RT-PCR confirmed RSV A and/or RSV B LRTD episodes at specified timepoints were included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | RSV_1_dose Group | RSV_annual Group
Number analyzed (Participants) | 107 | 22 | 22
Participants
  Nasal Congestion | 90 | 20 | 15
  Rhinorrhea | 96 | 20 | 19
  Sore Throat | 79 | 17 | 15
  Cough (new or increased) | 106 | 21 | 20
  Sputum (new or increased) | 95 | 19 | 17
  Shortness of breath or dyspnea (new or increased): number analyzed (Participants) | 106 | 22 | 22
  Shortness of breath or dyspnea (new or increased) | 72 | 14 | 13
  Wheezing (new or increased): number analyzed (Participants) | 106 | 22 | 22
  Wheezing (new or increased) | 56 | 15 | 10
  Crackles: number analyzed (Participants) | 100 | 22 | 21
  Crackles | 19 | 2 | 3
  Rhonchi: number analyzed (Participants) | 100 | 22 | 21
  Rhonchi | 31 | 5 | 7
  Respiratory rate ≥20 breaths/minute: number analyzed (Participants) | 103 | 22 | 22
  Respiratory rate ≥20 breaths/minute | 21 | 5 | 0
  Low or decreased oxygen saturation: number analyzed (Participants) | 103 | 22 | 22
  Low or decreased oxygen saturation | 8 | 1 | 4
  Fever: number analyzed (Participants) | 106 | 20 | 22
  Fever | 13 | 3 | 3
  Feverishness: number analyzed (Participants) | 107 | 21 | 22
  Feverishness | 44 | 7 | 8
  Fatigue | 86 | 16 | 15
  Body aches | 53 | 15 | 11
  Headache | 70 | 17 | 14
  Decreased appetite | 47 | 13 | 11
  Need for oxygen supplementation | 1 | 1 | 0
  Need for positive airway pressure therapy: number analyzed (Participants) | 106 | 22 | 22
  Need for positive airway pressure therapy | 0 | 1 | 0
  Need of other types of mechanical ventilation | 0 | 0 | 0
  Other symptoms or signs: number analyzed (Participants) | 106 | 22 | 22
  Other symptoms or signs | 28 | 3 | 5

31. Secondary Outcome: Number of Participants With Each Reported Symptom/Sign and Supportive Therapy Use Associated With of RT-PCR Confirmed RSV A and/or B LRTD Episodes During Season 3
Description: as for outcome 29
Time Frame: From start of Season 3 up to end of Season 3 in NH (a median of approximately 7 months)
Population: Analysis was performed on the mES-Dose 2. Only participants with data available for symptoms/signs and supportive therapy use associated with RT-PCR confirmed RSV A and/or RSV B LRTD episodes at specified timepoints were included in analysis. Only participants in NH were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | RSV_1_dose Group | RSV_annual Group
Number analyzed (Participants) | 61 | 16 | 6
Participants
  Nasal Congestion | 54 | 13 | 4
  Rhinorrhea | 50 | 14 | 4
  Sore Throat | 42 | 9 | 5
  Cough (new or increased) | 60 | 15 | 6
  Sputum (new or increased) | 53 | 14 | 5
  Shortness of breath or dyspnea (new or increased) | 38 | 9 | 4
  Wheezing (new or increased) | 32 | 5 | 3
  Crackles | 10 | 2 | 0
  Rhonchi | 16 | 8 | 2
  Respiratory rate ≥20 breaths/minute | 9 | 3 | 0
  Low or decreased oxygen saturation | 11 | 1 | 3
  Fever | 6 | 0 | 0
  Feverishness | 22 | 8 | 3
  Fatigue | 49 | 13 | 6
  Body aches | 39 | 10 | 5
  Headache | 41 | 10 | 5
  Decreased appetite | 33 | 11 | 3
  Need for oxygen supplementation | 0 | 1 | 0
  Need for positive airway pressure therapy | 0 | 0 | 0
  Need of other types of mechanical ventilation | 0 | 0 | 0
  Other symptoms or signs | 22 | 4 | 3

32. Secondary Outcome: Number of Participants With RT-PCR Confirmed RSV A and/or B ARI and LRTD Episodes According to Severity
Description: RSV A and/or B ARI and LRTD episodes were assessed as "mild", "moderate" or "severe" by the investigator after the single dose and after annual revaccination. Mild = an ARI/LRTD episode which is easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities. Moderate = an ARI/LRTD episode which is sufficiently discomforting to interfere with normal everyday activities. Severe = an ARI/LRTD episode which prevents normal, everyday activities.
Time Frame: Assessed during the study period (approximately 3 years for NH and 2.5-3 years for SH)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF3 Group | Placebo Group
Number analyzed (Participants) | 12468 | 12498
Participants
  Mild (Single dose) | 16 | 49
  Moderate (Single dose) | 29 | 138
  Severe (Single dose) | 3 | 28
  Mild (Annual revaccination) | 15 | 48
  Moderate (Annual revaccination) | 23 | 120
  Severe (Annual revaccination) | 0 | 24

33. Secondary Outcome: RSVPreF3 Specific Immunoglobulin G(IgG) Antibody Concentrations
Description: The RSVPreF3 IgG antibody concentrations are expressed as geometric mean concentrations (GMCs) in ELISA units per milliliter (EU/mL).
Time Frame: At pre-dose 1 (Day 1), Day 31 post-dose 1, pre-season 2 (approximately 10-17 months post Day 1 in NH; 12-21 months post Day 1 in SH) and pre-season 3 (approximately 24-27 months post Day 1, only in NH)
Population: Analysis was performed in a subset of participants from the Per Protocol Set for immunogenicity (PPSi), which included participants who received at least the first dose of the study intervention, have post-vaccination immunogenicity data available, and did not meet protocol deviations that lead to exclusion. Only participants with data available at specified timepoints were included in analysis. Analysis is presented dose-wise after first dose administration and annual revaccinations.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Placebo Group | RSV_1_dose Group | RSV_annual Group
Number analyzed (Participants) | 878 | 441 | 431
EU/mL
  Pre-dose 1 at day 1 | 7090.2 [6783.4 to 7410.9] | 6956.5 [6505.2 to 7439.2] | 7101.1 [6640.7 to 7593.4]
  Post-dose 1 at day 31: number analyzed (Participants) | 834 | 420 | 414
  Post-dose 1 at day 31 | 7053.2 [6732.0 to 7389.8] | 89361.9 [83409.6 to 95738.9] | 93769.5 [87896.6 to 100034.8]
  Pre-Season 2: number analyzed (Participants) | 669 | 346 | 317
  Pre-Season 2 | 7594.8 [7203.9 to 8007.0] | 24103.6 [22366.8 to 25975.3] | 24523.8 [22748.7 to 26437.4]
  Pre-Season 3: number analyzed (Participants) | 517 | 274 | 249
  Pre-Season 3 | 8436.6 [7927.3 to 8978.7] | 21255.0 [19587.7 to 23064.2] | 28925.3 [26928.0 to 31070.7]

34. Secondary Outcome: RSV A Neutralizing Antibody Titers
Description: The RSV A neutralizing antibody titers are expressed as geometric mean titers (GMTs).
Time Frame: as for outcome 33
Population: Analysis was performed in a subset of participants from the PPSi. Only participants with data available at specified timepoints were included in analysis. Analysis is presented dose-wise after first dose administration and annual revaccinations.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Placebo Group | RSV_1_dose Group | RSV_annual Group
Number analyzed (Participants) | 878 | 441 | 431
Titers
  Pre-dose 1 at day 1 | 933.5 [881.8 to 988.4] | 899.8 [829.1 to 976.5] | 929.3 [852.6 to 1013.0]
  Post-dose 1 at day 31: number analyzed (Participants) | 834 | 420 | 414
  Post-dose 1 at day 31 | 880.8 [828.9 to 935.9] | 8915.5 [8080.6 to 9836.8] | 9652.4 [8727.5 to 10675.3]
  Pre-Season 2: number analyzed (Participants) | 667 | 345 | 317
  Pre-Season 2 | 865.8 [809.6 to 925.9] | 2535.9 [2284.7 to 2814.8] | 2918.4 [2594.5 to 3282.9]
  Pre-Season 3: number analyzed (Participants) | 517 | 274 | 249
  Pre-Season 3 | 977.9 [905.5 to 1056.0] | 2049.7 [1841.0 to 2282.1] | 2996.1 [2665.3 to 3368.1]

35. Secondary Outcome: RSV B Neutralizing Antibody Titers
Description: RSV B neutralizing antibodies are expressed as GMTs.
Time Frame: as for outcome 33
Population: Analysis was performed on PPSi. Only participants with data available at specified timepoints were included in analysis. Analysis is presented dose-wise after first dose administration and annual revaccinations.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Placebo Group | RSV_1_dose Group | RSV_annual Group
Number analyzed (Participants) | 878 | 441 | 431
Titers
  Pre-dose 1 at day 1 | 1249.7 [1179.1 to 1324.5] | 1189.9 [1097.4 to 1290.2] | 1187.2 [1096.7 to 1285.2]
  Post-dose 1 at day 31: number analyzed (Participants) | 834 | 420 | 414
  Post-dose 1 at day 31 | 1262.4 [1183.8 to 1346.2] | 9928.9 [9103.7 to 10829.0] | 10253.4 [9362.7 to 11228.9]
  Pre-Season 2: number analyzed (Participants) | 667 | 346 | 317
  Pre-Season 2 | 1229.7 [1149.9 to 1315.1] | 2955.5 [2677.0 to 3262.9] | 2979.2 [2692.2 to 3296.9]
  Pre-Season 3: number analyzed (Participants) | 517 | 274 | 249
  Pre-Season 3 | 946.8 [873.5 to 1026.3] | 2054.5 [1829.9 to 2306.5] | 2515.3 [2249.9 to 2812.0]

36. Secondary Outcome: Number of Participants With Any and Grade 3 Solicited Administration Site Adverse Events
Description: Any solicited event is defined as the occurrence of any solicited adverse event (AE) regardless of intensity grade or relation to study vaccination. Grade 3 = an event which prevented normal, everyday activities. The assessed administration site events include pain, erythema and swelling.
Time Frame: During the 4-day follow up period after first vaccination (Day 1), second vaccination (administered pre-season 2) and after the third vaccination (administered pre-season 3 -only applicable for participants in NH])
Population: Analysis was performed on a subset of participants from the solicited safety set (SSS), which included participants who received at least the first dose of the study intervention and with the solicited administration site events diary card data available after the corresponding vaccination for the specified duration. Only participants with data available at specified timepoints were included in analysis. Analysis is presented dose-wise after first dose administration and annual revaccinations.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | RSV_1_dose Group | RSV_annual Group
Number analyzed (Participants) | 874 | 442 | 437
Participants
  Erythema, Dose 1, Any | 10 | 41 | 30
  Erythema, Dose 1, Grade 3 | 0 | 0 | 2
  Erythema, Dose 2, Any: number analyzed (Participants) | 657 | 341 | 323
  Erythema, Dose 2, Any | 1 | 1 | 31
  Erythema , Dose 2, Grade 3: number analyzed (Participants) | 657 | 341 | 323
  Erythema , Dose 2, Grade 3 | 0 | 0 | 3
  Erythema, Dose 3 (NH), Any: number analyzed (Participants) | 107 | 59 | 42
  Erythema, Dose 3 (NH), Any | 0 | 0 | 2
  Erythema, Dose 3 (NH), Grade 3: number analyzed (Participants) | 107 | 59 | 42
  Erythema, Dose 3 (NH), Grade 3 | 0 | 0 | 1
  Pain, Dose 1, Any | 81 | 267 | 268
  Pain, Dose 1, Grade 3 | 0 | 6 | 3
  Pain, Dose 2, Any: number analyzed (Participants) | 657 | 341 | 323
  Pain, Dose 2, Any | 51 | 30 | 169
  Pain, Dose 2, Grade 3: number analyzed (Participants) | 657 | 341 | 323
  Pain, Dose 2, Grade 3 | 0 | 0 | 2
  Pain, Dose 3 (NH), Any: number analyzed (Participants) | 107 | 59 | 42
  Pain, Dose 3 (NH), Any | 7 | 3 | 25
  Pain, Dose 3 (NH), Grade 3: number analyzed (Participants) | 107 | 59 | 42
  Pain, Dose 3 (NH), Grade 3 | 0 | 0 | 0
  Swelling, Dose 1, Any | 7 | 25 | 28
  Swelling, Dose 1, Grade 3 | 0 | 0 | 2
  Swelling, Dose 2, Any: number analyzed (Participants) | 657 | 341 | 323
  Swelling, Dose 2, Any | 2 | 0 | 23
  Swelling, Dose 2, Grade 3: number analyzed (Participants) | 657 | 341 | 323
  Swelling, Dose 2, Grade 3 | 0 | 0 | 6
  Swelling, Dose 3 (NH), Any: number analyzed (Participants) | 107 | 59 | 42
  Swelling, Dose 3 (NH), Any | 0 | 1 | 2
  Swelling, Dose 3 (NH), Grade 3: number analyzed (Participants) | 107 | 59 | 42
  Swelling, Dose 3 (NH), Grade 3 | 0 | 0 | 0

37. Secondary Outcome: Number of Participants With Any and Grade 3 Solicited Systemic Adverse Events
Description: Any solicited event is defined as the occurrence of any solicited adverse event (AE) regardless of intensity grade or relation to study vaccination. Grade 3 = an event which prevented normal, everyday activities. The assessed solicited systemic events include arthralgia, fatigue, fever, headache and myalgia. Fever is defined as a temperature ≥ 38.0°C by any route. Grade 3 fever is defined as temperature >39°C by any route.
Time Frame: as for outcome 36
Population: Analysis was performed on a subset of participants from the solicited safety set (SSS), which included participants who received at least the first dose of the study intervention and with the solicited systemic events diary card data available after the corresponding vaccination for the specified duration. Only participants with data available at specified timepoints were included in analysis. Analysis is presented dose-wise after first dose administration and annual revaccinations.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | RSV_1_dose Group | RSV_annual Group
Number analyzed (Participants) | 878 | 442 | 437
Participants
  Arthralgia, Dose 1, Any | 56 | 74 | 84
  Arthralgia, Dose 1, Grade 3 | 5 | 5 | 6
  Arthralgia, Dose 2, Any: number analyzed (Participants) | 656 | 341 | 323
  Arthralgia, Dose 2, Any | 48 | 20 | 55
  Arthralgia, Dose 2, Grade 3: number analyzed (Participants) | 656 | 341 | 323
  Arthralgia, Dose 2, Grade 3 | 2 | 0 | 2
  Arthralgia, Dose 3 (NH), Any: number analyzed (Participants) | 107 | 59 | 41
  Arthralgia, Dose 3 (NH), Any | 5 | 2 | 5
  Arthralgia, Dose 3 (NH), Grade 3: number analyzed (Participants) | 107 | 59 | 41
  Arthralgia, Dose 3 (NH), Grade 3 | 0 | 0 | 0
  Fatigue, Dose 1, Any | 141 | 143 | 153
  Fatigue, Dose 1, Grade 3 | 4 | 6 | 9
  Fatigue, Dose 2, Any: number analyzed (Participants) | 656 | 341 | 323
  Fatigue, Dose 2, Any | 80 | 44 | 98
  Fatigue, Dose 2, Grade 3: number analyzed (Participants) | 656 | 341 | 323
  Fatigue, Dose 2, Grade 3 | 7 | 2 | 3
  Fatigue, Dose 3 (NH), Any: number analyzed (Participants) | 107 | 59 | 41
  Fatigue, Dose 3 (NH), Any | 12 | 8 | 9
  Fatigue, Dose 3 (NH), Grade 3: number analyzed (Participants) | 107 | 59 | 41
  Fatigue, Dose 3 (NH), Grade 3 | 0 | 1 | 0
  Fever, Dose 1, Any | 3 | 14 | 4
  Fever, Dose 1, Grade 3 | 1 | 1 | 0
  Fever, Dose 2, Any: number analyzed (Participants) | 656 | 341 | 323
  Fever, Dose 2, Any | 4 | 1 | 6
  Fever, Dose 2, Grade 3: number analyzed (Participants) | 656 | 341 | 323
  Fever, Dose 2, Grade 3 | 2 | 0 | 0
  Fever, Dose 3 (NH), Any: number analyzed (Participants) | 107 | 59 | 41
  Fever, Dose 3 (NH), Any | 1 | 0 | 0
  Fever, Dose 3 (NH), Grade 3: number analyzed (Participants) | 107 | 59 | 41
  Fever, Dose 3 (NH), Grade 3 | 0 | 0 | 0
  Headache, Dose 1, Any | 111 | 116 | 123
  Headache, Dose 1, Grade 3 | 0 | 6 | 5
  Headache, Dose 2, Any: number analyzed (Participants) | 656 | 341 | 323
  Headache, Dose 2, Any | 60 | 41 | 73
  Headache, Dose 2, Grade 3: number analyzed (Participants) | 656 | 341 | 323
  Headache, Dose 2, Grade 3 | 4 | 1 | 2
  Headache, Dose 3 (NH), Any: number analyzed (Participants) | 107 | 59 | 41
  Headache, Dose 3 (NH), Any | 9 | 6 | 5
  Headache, Dose 3 (NH), Grade 3: number analyzed (Participants) | 107 | 59 | 41
  Headache, Dose 3 (NH), Grade 3 | 0 | 0 | 0
  Myalgia, Dose 1, Any | 72 | 127 | 128
  Myalgia, Dose 1, Grade 3 | 3 | 5 | 7
  Myalgia, Dose 2, Any: number analyzed (Participants) | 656 | 341 | 323
  Myalgia, Dose 2, Any | 52 | 20 | 82
  Myalgia, Dose 2, Grade 3: number analyzed (Participants) | 656 | 341 | 323
  Myalgia, Dose 2, Grade 3 | 3 | 0 | 3
  Myalgia, Dose 3 (NH), Any: number analyzed (Participants) | 107 | 59 | 41
  Myalgia, Dose 3 (NH), Any | 5 | 3 | 7
  Myalgia, Dose 3 (NH), Grade 3: number analyzed (Participants) | 107 | 59 | 41
  Myalgia, Dose 3 (NH), Grade 3 | 0 | 0 | 0

38. Secondary Outcome: Number of Days With Solicited Administration Site Adverse Events
Time Frame: as for outcome 36
Population: as for outcome 36
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo Group | RSV_1_dose Group | RSV_annual Group
Number analyzed (Participants) | 81 | 267 | 268
Days
  Erythema, Dose 1: number analyzed (Participants) | 10 | 41 | 30
  Erythema, Dose 1 | 4.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0]
  Erythema, Dose 2: number analyzed (Participants) | 1 | 1 | 31
  Erythema, Dose 2 | 4.0 [4.0 to 4.0] | 2.0 [2.0 to 2.0] | 3.0 [2.0 to 3.0]
  Erythema, Dose 3 (NH): number analyzed (Participants) | 0 | 0 | 2
  Erythema, Dose 3 (NH) |  |  | 3.0 [2.0 to 4.0]
  Pain, Dose 1 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0] | 2.0 [2.0 to 3.0]
  Pain, Dose 2: number analyzed (Participants) | 51 | 30 | 169
  Pain, Dose 2 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 2.0 [2.0 to 3.0]
  Pain, Dose 3 (NH): number analyzed (Participants) | 7 | 3 | 25
  Pain, Dose 3 (NH) | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0]
  Swelling, Dose 1: number analyzed (Participants) | 7 | 25 | 28
  Swelling, Dose 1 | 4.0 [2.0 to 8.0] | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.5]
  Swelling, Dose 2: number analyzed (Participants) | 2 | 0 | 23
  Swelling, Dose 2 | 2.0 [1.0 to 3.0] |  | 3.0 [2.0 to 4.0]
  Swelling, Dose 3 (NH): number analyzed (Participants) | 0 | 1 | 2
  Swelling, Dose 3 (NH) |  | 49.0 [49.0 to 49.0] | 1.5 [1.0 to 2.0]

39. Secondary Outcome: Number of Days With Solicited Systemic Adverse Events
Time Frame: as for outcome 36
Population: as for outcome 37
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo Group | RSV_1_dose Group | RSV_annual Group
Number analyzed (Participants) | 141 | 143 | 153
Days
  Arthralgia, Dose 1: number analyzed (Participants) | 56 | 74 | 84
  Arthralgia, Dose 1 | 2.5 [1.0 to 4.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Arthralgia, Dose 2: number analyzed (Participants) | 48 | 20 | 55
  Arthralgia, Dose 2 | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 3.0]
  Arthralgia, Dose 3 (NH): number analyzed (Participants) | 5 | 2 | 5
  Arthralgia, Dose 3 (NH) | 4.0 [3.0 to 4.0] | 2.0 [1.0 to 3.0] | 4.0 [1.0 to 4.0]
  Fatigue, Dose 1 | 1.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Fatigue, Dose 2: number analyzed (Participants) | 80 | 44 | 98
  Fatigue, Dose 2 | 2.0 [1.0 to 4.0] | 1.5 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Fatigue, Dose 3 (NH): number analyzed (Participants) | 12 | 8 | 9
  Fatigue, Dose 3 (NH) | 1.0 [1.0 to 2.0] | 2.5 [1.0 to 3.5] | 2.0 [1.0 to 2.0]
  Fever, Dose 1: number analyzed (Participants) | 3 | 14 | 4
  Fever, Dose 1 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.5]
  Fever, Dose 2: number analyzed (Participants) | 4 | 1 | 6
  Fever, Dose 2 | 2.0 [1.5 to 3.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 4.0]
  Fever, Dose 3 (NH): number analyzed (Participants) | 1 | 0 | 0
  Fever, Dose 3 (NH) | 1.0 [1.0 to 1.0] |  |
  Headache, Dose 1: number analyzed (Participants) | 111 | 116 | 123
  Headache, Dose 1 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Headache, Dose 2: number analyzed (Participants) | 60 | 41 | 73
  Headache, Dose 2 | 2.0 [1.0 to 4.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Headache, Dose 3 (NH): number analyzed (Participants) | 9 | 6 | 5
  Headache, Dose 3 (NH) | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0] | 2.0 [2.0 to 2.0]
  Myalgia, Dose 1: number analyzed (Participants) | 72 | 127 | 128
  Myalgia, Dose 1 | 1.5 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Myalgia, Dose 2: number analyzed (Participants) | 52 | 20 | 82
  Myalgia, Dose 2 | 2.0 [1.0 to 4.0] | 1.5 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Myalgia, Dose 3 (NH): number analyzed (Participants) | 5 | 3 | 7
  Myalgia, Dose 3 (NH) | 2.0 [1.0 to 3.0] | 3.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0]

40. Secondary Outcome: Number of Participants With Any Unsolicited AEs
Description: An unsolicited AE is defined as any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside of the specified period of follow-up for solicited symptoms was reported as an unsolicited AE. Any= occurrence of the event regardless of intensity grade or relation to the study vaccination.
Time Frame: During the 30-day follow up period after first vaccination (Day 1), second vaccination (administered pre-season 2) and after the third vaccination (administered pre-season 3 -only applicable for participants in NH)
Population: Analysis is performed on the Exposed Set, which included all participants that received at least the first vaccination. Only participants with data available at specified timepoints were included in analysis. Analysis is presented dose-wise after first dose administration and annual revaccinations.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | RSV_1_dose Group | RSV_annual Group
Number analyzed (Participants) | 12503 | 6226 | 6243
Participants
  Any unsolicited AE (post Dose 1) | 2334 | 2149 | 2136
  Any unsolicited AE (post Dose 2): number analyzed (Participants) | 10033 | 4988 | 4968
  Any unsolicited AE (post Dose 2) | 1570 | 824 | 1456
  Any unsolicited AE (post Dose 3): number analyzed (Participants) | 2866 | 1467 | 1409
  Any unsolicited AE (post Dose 3) | 422 | 233 | 397

41. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An SAE is defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect in the offspring of a study participant, or in other situations that were considered serious per medical or scientific judgment. Any = occurrence of any SAE regardless of intensity grade or relation to study vaccination.
Time Frame: From the day of the vaccination up to 6 months after each vaccination (first vaccination: at Day 1, second vaccination: at pre-season 2 and the third vaccination: at pre-season 3 -only applicable for participants in NH])
Population: as for outcome 40
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | RSV_1_dose Group | RSV_annual Group
Number analyzed (Participants) | 12503 | 6226 | 6243
Participants
  Any SAE (post Dose 1) | 541 | 280 | 268
  Any SAE (post Dose 2): number analyzed (Participants) | 10033 | 4988 | 4968
  Any SAE (post Dose 2) | 497 | 239 | 229
  Any SAE (post Dose 3): number analyzed (Participants) | 2866 | 1467 | 1409
  Any SAE (post Dose 3) | 179 | 75 | 73

42. Secondary Outcome: Number of Participants With Potential Immune Mediated Diseases (pIMDs)
Description: pIMDs aredefined as a subset of Adverse Events of Specific Interest (AESIs) that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology. Any= occurrence of any pIMD regardless of intensity grade or relation to the study vaccination.
Time Frame: as for outcome 41
Population: as for outcome 40
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | RSV_1_dose Group | RSV_annual Group
Number analyzed (Participants) | 12503 | 6226 | 6243
Participants
  Any pIMDs (post Dose 1) | 39 | 27 | 19
  Any pIMDs (post Dose 2): number analyzed (Participants) | 10033 | 4988 | 4968
  Any pIMDs (post Dose 2) | 39 | 19 | 14
  Any pIMDs (post Dose 3): number analyzed (Participants) | 2866 | 1467 | 1409
  Any pIMDs (post Dose 3) | 13 | 8 | 10

43. Secondary Outcome: Number of Participants With Related SAEs
Description: Related SAEs that occur throughout the study are assessed. Related SAEs= Any SAE related to investigational vaccine or related to study participation or to a GSK concomitant medication/vaccine as assessed by the investigator.
Time Frame: From Day 1 up to study end (approximately 3 years for NH and 2.5-3 years for SH)
Population: Analysis was performed on the Exposed Set. Only participants with data available at specified timepoints were included in analysis. Analysis is presented dose-wise after first dose administration and annual revaccinations.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | RSV_1_dose Group | RSV_annual Group
Number analyzed (Participants) | 12503 | 6226 | 6243
Participants | 12 | 8 | 12

44. Secondary Outcome: Number of Participants With Fatal SAEs
Description: Fatal SAEs that occur throughout the study are assessed. Fatal SAEs= Any SAEs leading to deaths.
Time Frame: From Day 1 up to study end (approximately 3 years for NH and 2.5-3 years for SH)
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | RSV_1_dose Group | RSV_annual Group
Number analyzed (Participants) | 12503 | 6226 | 6243
Participants | 265 | 111 | 120

45. Secondary Outcome: Number of Participants With Related pIMDs
Description: Related pIMD = pIMD assessed by the investigator as related to the study vaccination.
Time Frame: From Day 1 up to study end (approximately 3 years for NH and 2.5-3 years for SH)
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | RSV_1_dose Group | RSV_annual Group
Number analyzed (Participants) | 12503 | 6226 | 6243
Participants | 9 | 7 | 5

ADVERSE EVENTS:
Time Frame: Solicited AEs: during the 4-day follow-up period after any vaccination and unsolicited AEs: during the 30-day follow-up period after any vaccination. SAEs and pIMDs from Day 1 up to 6 months after any vaccination. All cause mortality, Fatal SAEs, Related SAEs and Related pIMDs were collected throughout the study period (From Day 1 up to approximately 3 years for NH and 2.5-3 years for SH)
Description: All adverse events are presented for the Exposed set, which included all participants that received at least one study intervention.
Groups:
- Placebo Group: Participants received 1 dose of placebo at Day 1 and an additional dose of placebo every subsequent year.
Arm/Group | Placebo Group | RSV_1_dose Group | RSV_annual Group
All-Cause Mortality (participants affected / at risk) | 265/12503 | 111/6226 | 120/6243
Serious Adverse Events (participants affected / at risk) | 1660/12503 | 799/6226 | 796/6243
Other Adverse Events (participants affected / at risk) | 5837/12503 | 3663/6226 | 3826/6243
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Group (N=12503) | RSV_1_dose Group (N=6226) | RSV_annual Group (N=6243)
Pneumonia (Infections and infestations) | 80 (84) | 37 (42) | 34 (35)
COVID-19 (Infections and infestations) | 34 (34) | 21 (21) | 19 (19)
COVID-19 pneumonia (Infections and infestations) | 26 (26) | 15 (15) | 14 (15)
Sepsis (Infections and infestations) | 22 (22) | 9 (9) | 13 (13)
Urinary tract infection (Infections and infestations) | 17 (17) | 9 (10) | 11 (12)
Cellulitis (Infections and infestations) | 12 (12) | 5 (5) | 5 (7)
Diverticulitis (Infections and infestations) | 9 (10) | 5 (5) | 4 (5)
Urosepsis (Infections and infestations) | 7 (7) | 4 (4) | 7 (7)
Lower respiratory tract infection (Infections and infestations) | 5 (5) | 7 (7) | 5 (5)
Appendicitis (Infections and infestations) | 5 (5) | 5 (5) | 6 (6)
Gastroenteritis (Infections and infestations) | 4 (4) | 8 (8) | 2 (2)
Bronchitis (Infections and infestations) | 7 (7) | 2 (2) | 4 (4)
Septic shock (Infections and infestations) | 5 (5) | 5 (5) | 3 (3)
Influenza (Infections and infestations) | 7 (7) | 1 (1) | 4 (4)
Osteomyelitis (Infections and infestations) | 7 (9) | 2 (2) | 3 (3)
Kidney infection (Infections and infestations) | 6 (6) | 3 (3) | 1 (1)
Pyelonephritis (Infections and infestations) | 4 (4) | 0 (0) | 5 (5)
Localised infection (Infections and infestations) | 6 (7) | 1 (1) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 4 (4) | 1 (1) | 3 (4)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 6 (6) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 5 (5) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 2 (2) | 2 (2) | 2 (2)
Erysipelas (Infections and infestations) | 1 (1) | 1 (1) | 4 (6)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 2 (2) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
Wound infection (Infections and infestations) | 3 (3) | 1 (1) | 2 (2)
Arthritis bacterial (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Escherichia sepsis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Post procedural infection (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Arthritis infective (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Device related infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Diabetic foot infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Epididymitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Liver abscess (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Abdominal sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Atypical mycobacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bursitis infective (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Colonic abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Diverticulitis intestinal perforated (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Gangrene (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Groin abscess (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Nosocomial infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Psoas abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Spinal cord infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Blister infected (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Candida pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Capnocytophaga sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cardiac valve vegetation (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Coccidioidomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Endocarditis staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Extradural abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gallbladder empyema (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer helicobacter (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Giardiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatitis E (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Human anaplasmosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Incision site abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infective aortitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infective exacerbation of asthma (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Joint abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Neurosyphilis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post-acute COVID-19 syndrome (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postoperative abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Renal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory moniliasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rotavirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Scrotal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Scrotal cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Scrotal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Submandibular abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Toxic shock syndrome streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 66 (77) | 22 (22) | 31 (35)
Myocardial infarction (Cardiac disorders) | 54 (56) | 17 (18) | 16 (16)
Coronary artery disease (Cardiac disorders) | 37 (38) | 7 (8) | 18 (20)
Acute myocardial infarction (Cardiac disorders) | 27 (27) | 13 (13) | 15 (16)
Cardiac failure (Cardiac disorders) | 29 (34) | 12 (14) | 14 (15)
Cardiac failure congestive (Cardiac disorders) | 20 (21) | 14 (14) | 10 (10)
Angina pectoris (Cardiac disorders) | 10 (10) | 8 (8) | 7 (7)
Angina unstable (Cardiac disorders) | 16 (17) | 3 (3) | 5 (5)
Cardiac arrest (Cardiac disorders) | 14 (15) | 6 (6) | 4 (5)
Myocardial ischaemia (Cardiac disorders) | 13 (14) | 2 (2) | 6 (6)
Atrial flutter (Cardiac disorders) | 6 (6) | 6 (6) | 6 (8)
Arteriosclerosis coronary artery (Cardiac disorders) | 4 (4) | 3 (3) | 4 (4)
Acute coronary syndrome (Cardiac disorders) | 4 (4) | 5 (6) | 1 (1)
Arrhythmia (Cardiac disorders) | 6 (6) | 3 (3) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 6 (6) | 3 (3) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 3 (3) | 2 (2) | 4 (4)
Aortic valve stenosis (Cardiac disorders) | 5 (5) | 3 (3) | 0 (0)
Bradycardia (Cardiac disorders) | 6 (6) | 2 (2) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 5 (5) | 1 (1) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 3 (3) | 4 (4) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 3 (3) | 1 (1) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 3 (3) | 3 (4) | 0 (0)
Left ventricular failure (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1)
Pericarditis (Cardiac disorders) | 4 (4) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 3 (3) | 0 (0) | 3 (3)
Atrioventricular block complete (Cardiac disorders) | 3 (3) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 3 (3) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 3 (3) | 1 (1) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 4 (4) | 0 (0) | 0 (0)
Dilated cardiomyopathy (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Heart failure with reduced ejection fraction (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 2 (3) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Aortic valve disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiomegaly (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiorenal syndrome (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Chronic coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Chordae tendinae rupture (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery aneurysm (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery embolism (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Dressler's syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Heart failure with preserved ejection fraction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Mitral valve calcification (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Nodal rhythm (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Paroxysmal atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 39 (39) | 20 (20) | 15 (15)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21 (21) | 10 (10) | 10 (10)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (13) | 7 (7) | 7 (7)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 9 (10) | 5 (5)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 6 (6) | 3 (3)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 4 (4) | 4 (4)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4) | 4 (4)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4) | 2 (2)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 4 (4)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (1) | 2 (2)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 1 (1) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1) | 2 (2)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1) | 2 (3)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 2 (2)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 3 (3)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 2 (2)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 4 (4)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 0 (0) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 2 (2)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (4) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Paget's disease of nipple (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bile duct adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Borderline ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Breast cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Endometrial cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Endometrial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Fallopian tube neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Follicular lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Gastrointestinal lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Head and neck cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hepatic cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hypopharyngeal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Intraductal papillary-mucinous carcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to chest wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to rectum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastatic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Myxoid liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Non-small cell lung cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pseudomyxoma peritonei (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Soft tissue sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of the hypopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 46 (47) | 15 (15) | 22 (22)
Syncope (Nervous system disorders) | 21 (21) | 22 (22) | 13 (13)
Transient ischaemic attack (Nervous system disorders) | 26 (27) | 7 (7) | 10 (10)
Ischaemic stroke (Nervous system disorders) | 8 (8) | 6 (6) | 7 (7)
Cerebral haemorrhage (Nervous system disorders) | 7 (7) | 4 (4) | 5 (5)
Dizziness (Nervous system disorders) | 4 (4) | 6 (7) | 3 (4)
Subarachnoid haemorrhage (Nervous system disorders) | 8 (8) | 1 (1) | 3 (3)
Carotid artery stenosis (Nervous system disorders) | 4 (4) | 2 (2) | 3 (3)
Loss of consciousness (Nervous system disorders) | 4 (4) | 2 (2) | 3 (3)
Seizure (Nervous system disorders) | 2 (2) | 3 (3) | 3 (3)
Sciatica (Nervous system disorders) | 3 (3) | 1 (1) | 3 (3)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2)
Cerebral infarction (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 3 (4) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Transient global amnesia (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Brain injury (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Cerebral arteriosclerosis (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Cerebellar stroke (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Facial paresis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Arachnoiditis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Brain stem haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Brain stem stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebellar haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebellar syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral venous sinus thrombosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrospinal fistula (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cervical cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Demyelinating polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Diplegia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dural arteriovenous fistula (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Intracranial haematoma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lacunar stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbosacral radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Mental impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Myelin oligodendrocyte glycoprotein antibody-associated disease (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuroleptic malignant syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Occipital lobe stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Occipital neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Psychogenic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Senile dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal claudication (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Thalamus haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Thoracic radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombotic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vertebral artery occlusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vertebrobasilar artery dissection (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vertebrobasilar stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 17 (17) | 8 (8) | 9 (10)
Hip fracture (Injury, poisoning and procedural complications) | 14 (14) | 9 (9) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 10 (10) | 7 (7) | 5 (5)
Rib fracture (Injury, poisoning and procedural complications) | 11 (11) | 4 (4) | 4 (4)
Ankle fracture (Injury, poisoning and procedural complications) | 10 (10) | 4 (4) | 3 (3)
Femoral neck fracture (Injury, poisoning and procedural complications) | 8 (8) | 5 (5) | 4 (4)
Pelvic fracture (Injury, poisoning and procedural complications) | 5 (5) | 3 (3) | 5 (5)
Radius fracture (Injury, poisoning and procedural complications) | 9 (9) | 2 (2) | 2 (2)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 5 (5) | 4 (4) | 2 (2)
Tendon rupture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 5 (5)
Joint dislocation (Injury, poisoning and procedural complications) | 5 (5) | 0 (0) | 3 (3)
Road traffic accident (Injury, poisoning and procedural complications) | 5 (5) | 2 (2) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 7 (7) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 3 (3)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 3 (3)
Humerus fracture (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 3 (3)
Incisional hernia (Injury, poisoning and procedural complications) | 4 (4) | 3 (3) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 2 (2)
Lower limb fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 2 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 3 (3)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Shoulder fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Post procedural hypotension (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Craniofacial fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Craniofacial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Flail chest (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hypobarism (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ilium fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Kidney rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative hypertension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radiation injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal cord injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Splenic injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Traumatic arthrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Trunk injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ulnar nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Urinary tract procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 13 (13) | 5 (5) | 8 (8)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 (9) | 4 (4) | 4 (4)
Intestinal obstruction (Gastrointestinal disorders) | 7 (7) | 7 (7) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 5 (5) | 6 (6) | 5 (5)
Gastritis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 7 (8)
Large intestine polyp (Gastrointestinal disorders) | 5 (5) | 1 (1) | 3 (3)
Colitis (Gastrointestinal disorders) | 5 (5) | 0 (0) | 3 (3)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (3)
Umbilical hernia (Gastrointestinal disorders) | 6 (6) | 0 (0) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (6) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 1 (1) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3)
Pancreatitis acute (Gastrointestinal disorders) | 4 (4) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 0 (0) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pancreatitis necrotising (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Peptic ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Appendix disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Coeliac artery compression syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epiploic appendagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oedematous pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal mucosal tear (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatic failure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Strangulated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Superior mesenteric artery syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 38 (53) | 24 (28) | 18 (23)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 31 (31) | 6 (6) | 15 (15)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 5 (6) | 6 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 5 (5) | 5 (5)
Asthma (Respiratory, thoracic and mediastinal disorders) | 8 (12) | 3 (3) | 6 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 4 (5) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 3 (3) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 1 (1) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma late onset (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Laryngeal polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lung perforation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Middle lobe syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 48 (52) | 38 (41) | 21 (21)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (2) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (4) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 3 (3)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 2 (2)
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff tear arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 54 (54) | 18 (18) | 28 (28)
Chest pain (General disorders) | 17 (17) | 11 (11) | 13 (13)
Multiple organ dysfunction syndrome (General disorders) | 6 (6) | 2 (2) | 2 (2)
Asthenia (General disorders) | 8 (8) | 0 (0) | 1 (1)
Sudden death (General disorders) | 6 (6) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 5 (5) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 2 (2) | 1 (1)
Sudden cardiac death (General disorders) | 2 (2) | 1 (1) | 1 (1)
Impaired healing (General disorders) | 3 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 1 (1)
Accidental death (General disorders) | 2 (2) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiac death (General disorders) | 2 (2) | 0 (0) | 0 (0)
Cyst rupture (General disorders) | 0 (0) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 0 (0)
Oedema (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 1 (1) | 0 (0)
Drowning (General disorders) | 1 (1) | 0 (0) | 0 (0)
Drug resistance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gait inability (General disorders) | 0 (0) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Ill-defined disorder (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Nodule (General disorders) | 0 (0) | 0 (0) | 1 (1)
Obstruction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic mass (General disorders) | 1 (1) | 0 (0) | 0 (0)
Stenosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Swelling face (General disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular stent occlusion (General disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 11 (11) | 7 (9) | 3 (3)
Hypertension (Vascular disorders) | 11 (11) | 0 (0) | 5 (5)
Aortic stenosis (Vascular disorders) | 3 (3) | 4 (4) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 5 (5) | 0 (0) | 4 (4)
Peripheral ischaemia (Vascular disorders) | 5 (5) | 3 (3) | 1 (1)
Hypertensive crisis (Vascular disorders) | 3 (3) | 2 (2) | 2 (2)
Hypotension (Vascular disorders) | 3 (3) | 2 (2) | 2 (2)
Circulatory collapse (Vascular disorders) | 4 (4) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 4 (4) | 1 (1) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 2 (2) | 2 (2)
Giant cell arteritis (Vascular disorders) | 2 (2) | 0 (0) | 3 (3)
Aortic aneurysm rupture (Vascular disorders) | 4 (4) | 0 (0) | 0 (0)
Extremity necrosis (Vascular disorders) | 2 (2) | 2 (2) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
Aortic dissection (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
Peripheral venous disease (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Aneurysm ruptured (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hypertensive urgency (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Internal haemorrhage (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Shock haemorrhagic (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Accelerated hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Aneurysm (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Arterial rupture (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Femoral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Iliac artery stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Malignant hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Scalp haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Subclavian steal syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 18 (19) | 12 (12) | 14 (14)
Nephrolithiasis (Renal and urinary disorders) | 8 (8) | 5 (5) | 7 (7)
Renal failure (Renal and urinary disorders) | 5 (5) | 2 (2) | 3 (3)
Ureterolithiasis (Renal and urinary disorders) | 6 (6) | 2 (2) | 1 (1)
Urinary retention (Renal and urinary disorders) | 8 (8) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 1 (1) | 3 (3)
Haematuria (Renal and urinary disorders) | 4 (4) | 2 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 3 (3) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Haemorrhage urinary tract (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Bladder disorder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder tamponade (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Obstructive nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureteral necrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (6) | 4 (4) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (7) | 3 (3) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (6) | 1 (1) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 6 (6) | 2 (2) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Diabetic complication (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Euglycaemic diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperchloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 21 (21) | 4 (4) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 9 (9) | 4 (4) | 3 (3)
Cholecystitis acute (Hepatobiliary disorders) | 8 (8) | 3 (3) | 5 (5)
Bile duct stone (Hepatobiliary disorders) | 4 (4) | 0 (0) | 2 (2)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 2 (2) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 2 (2)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 2 (2)
Biliary tract disorder (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 2 (4) | 0 (0) | 0 (0)
Gallbladder rupture (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Biliary dilatation (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis obstructive (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic haemorrhage (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 8 (8) | 4 (4) | 4 (4)
Confusional state (Psychiatric disorders) | 5 (5) | 1 (1) | 2 (3)
Mental status changes (Psychiatric disorders) | 5 (5) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 3 (4) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1)
Suicide attempt (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Completed suicide (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Mental disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Conversion disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Gender dysphoria (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hallucinations, mixed (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Substance-induced mood disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 13 (13) | 4 (4) | 4 (4)
Prostatitis (Reproductive system and breast disorders) | 4 (4) | 2 (2) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 2 (2)
Prostatomegaly (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0)
Genital prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
Adnexa uteri cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Breast hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic organ prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatic cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Prostatic dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Rectocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Scrotal swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 14 (15) | 6 (7) | 10 (12)
Glaucoma (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Ocular myasthenia (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Blepharochalasis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Blindness (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Blindness transient (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Corneal decompensation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Corneal erosion (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Episcleritis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eyelid cyst (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Macular degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinoschisis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 12 (12) | 6 (6) | 6 (6)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 1 (1)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pemphigus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Superficial inflammatory dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 3 (3) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood electrolytes abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio fluctuation (Investigations) | 1 (1) | 0 (0) | 0 (0)
Myocardial necrosis marker increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Pulse absent (Investigations) | 0 (0) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 4 (4) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Adrenal mass (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Cushing's syndrome (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Pituitary-dependent Cushing's syndrome (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 3 (3) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Primary amyloidosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 1 (1) | 0 (0)
Corneal dystrophy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Hereditary haemorrhagic telangiectasia (Congenital, familial and genetic disorders) | 1 (2) | 0 (0) | 0 (0)
Hereditary non-polyposis colorectal cancer syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Neurosensory hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 1 (1) | 0 (0)
Device loosening (Product Issues) | 2 (2) | 0 (0) | 0 (0)
Device breakage (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Assisted suicide (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Group (N=12503) | RSV_1_dose Group (N=6226) | RSV_annual Group (N=6243)
Fatigue (General disorders) | 410 (469) | 394 (446) | 453 (541)
Injection site erythema (General disorders) | 56 (60) | 291 (299) | 449 (522)
Injection site swelling (General disorders) | 38 (38) | 208 (211) | 347 (406)
Pyrexia (General disorders) | 85 (89) | 144 (149) | 197 (217)
Pain (General disorders) | 76 (78) | 76 (76) | 120 (129)
Chills (General disorders) | 46 (51) | 45 (45) | 104 (113)
Vaccination site pain (General disorders) | 18 (20) | 66 (67) | 86 (95)
Injection site pruritus (General disorders) | 24 (24) | 41 (41) | 84 (90)
Malaise (General disorders) | 34 (37) | 35 (38) | 69 (73)
Asthenia (General disorders) | 36 (36) | 40 (41) | 55 (58)
Injection site warmth (General disorders) | 5 (5) | 41 (43) | 78 (85)
Injection site joint pain (General disorders) | 9 (9) | 37 (40) | 50 (52)
Administration site pain (General disorders) | 8 (9) | 29 (30) | 54 (64)
Injection site reaction (General disorders) | 13 (13) | 29 (30) | 39 (46)
Injection site bruising (General disorders) | 25 (25) | 17 (17) | 30 (30)
Chest pain (General disorders) | 27 (28) | 25 (25) | 15 (15)
Feeling hot (General disorders) | 12 (12) | 20 (20) | 33 (33)
Oedema peripheral (General disorders) | 27 (27) | 12 (12) | 15 (15)
Influenza like illness (General disorders) | 26 (26) | 11 (13) | 13 (13)
Injection site discomfort (General disorders) | 4 (4) | 12 (12) | 24 (25)
Peripheral swelling (General disorders) | 19 (19) | 11 (11) | 10 (10)
Injection site induration (General disorders) | 4 (4) | 12 (12) | 23 (23)
Vaccination site erythema (General disorders) | 2 (2) | 11 (11) | 23 (26)
Vaccination site swelling (General disorders) | 0 (0) | 12 (12) | 24 (27)
Chest discomfort (General disorders) | 13 (13) | 8 (8) | 10 (10)
Injection site oedema (General disorders) | 1 (1) | 5 (5) | 22 (24)
Feeling cold (General disorders) | 6 (7) | 9 (9) | 10 (11)
Injection site inflammation (General disorders) | 4 (4) | 7 (7) | 14 (14)
Injection site rash (General disorders) | 4 (4) | 10 (11) | 11 (11)
Discomfort (General disorders) | 5 (5) | 8 (8) | 11 (11)
Injection site haematoma (General disorders) | 10 (10) | 5 (5) | 7 (7)
Administration site erythema (General disorders) | 1 (1) | 6 (6) | 13 (14)
Swelling (General disorders) | 5 (5) | 7 (7) | 7 (7)
Axillary pain (General disorders) | 4 (4) | 4 (4) | 9 (9)
Cyst (General disorders) | 7 (7) | 4 (6) | 5 (5)
Injection site movement impairment (General disorders) | 1 (1) | 5 (5) | 9 (9)
Injection site mass (General disorders) | 3 (3) | 3 (3) | 8 (9)
Administration site swelling (General disorders) | 1 (1) | 4 (4) | 7 (7)
Vaccination site pruritus (General disorders) | 2 (2) | 3 (3) | 7 (7)
Injection site hypoaesthesia (General disorders) | 6 (6) | 2 (2) | 3 (3)
Vaccination site reaction (General disorders) | 2 (2) | 7 (7) | 2 (2)
Adverse drug reaction (General disorders) | 2 (2) | 4 (4) | 3 (3)
Non-cardiac chest pain (General disorders) | 5 (5) | 2 (2) | 2 (2)
Injection site hyperaesthesia (General disorders) | 1 (1) | 2 (2) | 5 (6)
Swelling face (General disorders) | 5 (5) | 1 (1) | 2 (2)
Feeling abnormal (General disorders) | 1 (1) | 1 (1) | 5 (5)
Injection site haemorrhage (General disorders) | 2 (2) | 2 (2) | 3 (3)
Vaccination site bruising (General disorders) | 3 (3) | 2 (2) | 2 (2)
Hernia (General disorders) | 1 (1) | 1 (1) | 4 (4)
Illness (General disorders) | 3 (3) | 2 (2) | 1 (1)
Inflammation (General disorders) | 1 (1) | 1 (1) | 4 (4)
Injection site hypersensitivity (General disorders) | 0 (0) | 2 (2) | 4 (4)
Injection site paraesthesia (General disorders) | 3 (3) | 2 (2) | 1 (1)
Vaccination site warmth (General disorders) | 0 (0) | 2 (2) | 4 (4)
Administration site warmth (General disorders) | 1 (1) | 1 (1) | 3 (3)
Gait disturbance (General disorders) | 2 (2) | 1 (1) | 2 (2)
Injection site lymphadenopathy (General disorders) | 0 (0) | 3 (3) | 2 (2)
Injection site nodule (General disorders) | 1 (1) | 3 (3) | 1 (1)
Oedema (General disorders) | 3 (3) | 1 (1) | 1 (1)
Temperature regulation disorder (General disorders) | 1 (1) | 1 (1) | 3 (3)
Vessel puncture site bruise (General disorders) | 2 (2) | 1 (1) | 2 (2)
Ill-defined disorder (General disorders) | 1 (1) | 2 (4) | 1 (1)
Injection site urticaria (General disorders) | 1 (1) | 2 (2) | 1 (1)
Administration site joint pain (General disorders) | 0 (0) | 0 (0) | 3 (3)
Facial pain (General disorders) | 1 (1) | 1 (1) | 1 (1)
Feeling of body temperature change (General disorders) | 1 (1) | 1 (1) | 1 (1)
Injection site extravasation (General disorders) | 1 (1) | 0 (0) | 2 (2)
Injection site irritation (General disorders) | 1 (1) | 2 (2) | 0 (0)
Mass (General disorders) | 2 (2) | 0 (0) | 1 (1)
Nodule (General disorders) | 3 (3) | 0 (0) | 0 (0)
Precancerous condition (General disorders) | 1 (1) | 1 (1) | 1 (1)
Puncture site erythema (General disorders) | 0 (0) | 1 (1) | 2 (2)
Puncture site pain (General disorders) | 1 (1) | 1 (1) | 1 (1)
Secretion discharge (General disorders) | 1 (1) | 1 (1) | 1 (1)
Thirst (General disorders) | 1 (1) | 1 (1) | 1 (1)
Vaccination site inflammation (General disorders) | 0 (0) | 2 (2) | 1 (1)
Vaccination site movement impairment (General disorders) | 0 (0) | 1 (1) | 2 (2)
Administration site bruise (General disorders) | 0 (0) | 0 (0) | 2 (2)
Administration site pruritus (General disorders) | 0 (0) | 0 (0) | 2 (2)
Calcinosis (General disorders) | 0 (0) | 0 (0) | 2 (2)
Complication associated with device (General disorders) | 1 (1) | 0 (0) | 1 (1)
Granuloma (General disorders) | 2 (3) | 0 (0) | 0 (0)
Gravitational oedema (General disorders) | 2 (2) | 0 (0) | 0 (0)
Injection site discolouration (General disorders) | 1 (1) | 0 (0) | 1 (1)
Injection site joint discomfort (General disorders) | 0 (0) | 2 (2) | 0 (0)
Sensation of foreign body (General disorders) | 0 (0) | 1 (1) | 1 (1)
Vaccination site discolouration (General disorders) | 1 (1) | 1 (1) | 0 (0)
Vaccination site discomfort (General disorders) | 2 (2) | 0 (0) | 0 (0)
Vaccination site haematoma (General disorders) | 1 (1) | 0 (0) | 1 (1)
Vaccination site rash (General disorders) | 1 (1) | 0 (0) | 1 (1)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Administration site papule (General disorders) | 0 (0) | 1 (1) | 0 (0)
Application site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Application site warmth (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic fatigue syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Drug intolerance (General disorders) | 0 (0) | 1 (1) | 0 (0)
Exercise tolerance decreased (General disorders) | 0 (0) | 1 (1) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fat necrosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fat tissue increased (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fibrosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site coldness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site dermatitis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site joint movement impairment (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site joint swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site scab (General disorders) | 1 (1) | 0 (0) | 0 (0)
Local reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Medical device pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Meteoropathy (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvic mass (General disorders) | 1 (1) | 0 (0) | 0 (0)
Puncture site swelling (General disorders) | 0 (0) | 0 (0) | 1 (2)
Sluggishness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Suprapubic pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Ulcer haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vaccination site joint pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vaccination site joint swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vaccination site mass (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vaccination site paraesthesia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Withdrawal syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1178 (1283) | 600 (656) | 601 (647)
Upper respiratory tract infection (Infections and infestations) | 526 (638) | 244 (288) | 243 (298)
Bronchitis (Infections and infestations) | 204 (220) | 126 (139) | 99 (103)
Urinary tract infection (Infections and infestations) | 184 (214) | 85 (95) | 92 (106)
Nasopharyngitis (Infections and infestations) | 178 (190) | 90 (96) | 89 (92)
Respiratory tract infection (Infections and infestations) | 93 (96) | 54 (59) | 53 (57)
Sinusitis (Infections and infestations) | 90 (97) | 42 (44) | 46 (51)
Lower respiratory tract infection (Infections and infestations) | 61 (66) | 24 (26) | 31 (35)
Rhinitis (Infections and infestations) | 52 (52) | 28 (33) | 30 (32)
Pneumonia (Infections and infestations) | 61 (62) | 29 (29) | 19 (20)
Viral upper respiratory tract infection (Infections and infestations) | 48 (55) | 28 (32) | 25 (35)
Herpes zoster (Infections and infestations) | 49 (52) | 17 (18) | 31 (32)
Cystitis (Infections and infestations) | 43 (45) | 23 (27) | 18 (19)
Gastroenteritis (Infections and infestations) | 36 (36) | 25 (25) | 14 (15)
Influenza (Infections and infestations) | 30 (31) | 20 (20) | 24 (25)
Cellulitis (Infections and infestations) | 34 (36) | 14 (15) | 17 (17)
Oral herpes (Infections and infestations) | 31 (31) | 17 (17) | 17 (19)
Conjunctivitis (Infections and infestations) | 33 (34) | 9 (9) | 19 (20)
Ear infection (Infections and infestations) | 29 (32) | 14 (16) | 13 (13)
Tooth infection (Infections and infestations) | 27 (27) | 16 (16) | 9 (9)
Tooth abscess (Infections and infestations) | 26 (27) | 12 (13) | 13 (13)
Diverticulitis (Infections and infestations) | 23 (25) | 11 (13) | 9 (10)
Pharyngitis (Infections and infestations) | 21 (21) | 14 (15) | 8 (8)
Respiratory tract infection viral (Infections and infestations) | 11 (11) | 11 (12) | 12 (12)
Localised infection (Infections and infestations) | 15 (15) | 9 (10) | 9 (9)
Acute sinusitis (Infections and infestations) | 13 (13) | 9 (9) | 8 (12)
Suspected COVID-19 (Infections and infestations) | 14 (14) | 7 (8) | 8 (8)
Gingivitis (Infections and infestations) | 10 (11) | 7 (7) | 9 (9)
Viral infection (Infections and infestations) | 12 (12) | 2 (2) | 10 (10)
Otitis media (Infections and infestations) | 10 (11) | 4 (4) | 9 (9)
Hordeolum (Infections and infestations) | 8 (8) | 8 (8) | 6 (6)
Laryngitis (Infections and infestations) | 9 (9) | 7 (7) | 6 (6)
Lower respiratory tract infection viral (Infections and infestations) | 9 (9) | 8 (8) | 5 (5)
Otitis externa (Infections and infestations) | 12 (12) | 4 (6) | 5 (5)
Gastroenteritis viral (Infections and infestations) | 10 (10) | 6 (6) | 4 (4)
Eye infection (Infections and infestations) | 6 (7) | 6 (6) | 5 (5)
Fungal infection (Infections and infestations) | 7 (7) | 3 (4) | 7 (7)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 8 (8) | 4 (4) | 4 (4)
Helicobacter infection (Infections and infestations) | 6 (6) | 1 (1) | 8 (8)
Kidney infection (Infections and infestations) | 7 (7) | 2 (2) | 6 (6)
COVID-19 pneumonia (Infections and infestations) | 8 (8) | 2 (2) | 4 (4)
Onychomycosis (Infections and infestations) | 7 (7) | 4 (4) | 3 (3)
Periodontitis (Infections and infestations) | 9 (9) | 4 (4) | 1 (1)
Herpes simplex (Infections and infestations) | 8 (9) | 4 (4) | 1 (1)
Paronychia (Infections and infestations) | 5 (5) | 4 (4) | 3 (3)
Skin infection (Infections and infestations) | 5 (5) | 2 (2) | 5 (6)
Candida infection (Infections and infestations) | 8 (8) | 0 (0) | 3 (3)
Erysipelas (Infections and infestations) | 5 (5) | 4 (6) | 2 (2)
Oral candidiasis (Infections and infestations) | 4 (4) | 3 (3) | 4 (4)
Vulvovaginal candidiasis (Infections and infestations) | 6 (6) | 2 (2) | 2 (2)
Wound infection (Infections and infestations) | 4 (4) | 5 (5) | 1 (2)
Lower respiratory tract infection bacterial (Infections and infestations) | 7 (7) | 1 (1) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 4 (4) | 2 (2) | 3 (3)
Post-acute COVID-19 syndrome (Infections and infestations) | 2 (2) | 4 (4) | 3 (3)
Tinea pedis (Infections and infestations) | 3 (4) | 1 (1) | 5 (5)
Chronic sinusitis (Infections and infestations) | 1 (1) | 3 (3) | 4 (4)
Lyme disease (Infections and infestations) | 3 (3) | 2 (2) | 3 (3)
Tracheobronchitis (Infections and infestations) | 2 (2) | 4 (4) | 2 (2)
Bronchitis viral (Infections and infestations) | 1 (1) | 3 (3) | 3 (3)
Fungal skin infection (Infections and infestations) | 5 (5) | 2 (2) | 0 (0)
Furuncle (Infections and infestations) | 3 (3) | 2 (2) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 4 (4) | 1 (1) | 2 (2)
Herpes virus infection (Infections and infestations) | 2 (2) | 1 (1) | 4 (4)
Infective exacerbation of asthma (Infections and infestations) | 3 (3) | 3 (3) | 1 (1)
Otitis media acute (Infections and infestations) | 3 (3) | 1 (1) | 3 (3)
Post procedural infection (Infections and infestations) | 2 (2) | 3 (3) | 2 (2)
Pulpitis dental (Infections and infestations) | 4 (5) | 2 (2) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 3 (3) | 3 (3) | 1 (1)
Rhinovirus infection (Infections and infestations) | 5 (5) | 1 (1) | 1 (1)
Acarodermatitis (Infections and infestations) | 3 (3) | 1 (1) | 2 (2)
Infected bite (Infections and infestations) | 2 (2) | 3 (3) | 1 (1)
Postoperative wound infection (Infections and infestations) | 4 (5) | 0 (0) | 2 (2)
Staphylococcal infection (Infections and infestations) | 3 (3) | 2 (2) | 1 (1)
Tonsillitis (Infections and infestations) | 3 (4) | 1 (1) | 2 (2)
Folliculitis (Infections and infestations) | 2 (2) | 0 (0) | 3 (4)
Nail infection (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
Tinea cruris (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1) | 4 (4)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Impetigo (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Infected dermal cyst (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Infected skin ulcer (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Vaginal infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Viral pharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Vulvitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Abscess oral (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Fungal foot infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Genital infection fungal (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Helicobacter gastritis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Infected cyst (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Latent tuberculosis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Nail bed infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Urethritis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Viral sinusitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Dermatophytosis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Dermatophytosis of nail (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Dientamoeba infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Dysentery (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Eczema infected (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Enterovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Fungal oesophagitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gastric infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Laryngitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Laryngopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Norovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 1 (2) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Otitis media chronic (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pertussis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Root canal infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Salmonellosis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Sialoadenitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Viral rhinitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Acariasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Campylobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Chlamydial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dental gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dermatitis infected (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterobiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Eyelid infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungal pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal bacterial overgrowth (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Genital infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gingival abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
HIV infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Haemophilus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoid infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpangina (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes ophthalmic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Histoplasmosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Injection site pustule (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Laryngitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lyme arthritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lymphangitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Mycoplasma infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Myiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasal vestibulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis externa fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Penile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Perineal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pilonidal disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postoperative abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Prostate infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyonephrosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Retinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rocky mountain spotted fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Scarlet fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sebaceous gland infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Shigella infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinobronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin graft infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 424 (469) | 1379 (1462) | 1713 (2257)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Stenotrophomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Superinfection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vulval abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 710 (856) | 594 (712) | 664 (820)
Dizziness (Nervous system disorders) | 105 (112) | 66 (73) | 88 (91)
Sciatica (Nervous system disorders) | 43 (44) | 18 (18) | 21 (21)
Lethargy (Nervous system disorders) | 14 (14) | 19 (21) | 13 (13)
Syncope (Nervous system disorders) | 20 (21) | 9 (9) | 12 (12)
Paraesthesia (Nervous system disorders) | 17 (17) | 13 (13) | 9 (9)
Migraine (Nervous system disorders) | 20 (25) | 6 (6) | 9 (12)
Hypoaesthesia (Nervous system disorders) | 12 (12) | 14 (15) | 8 (8)
Carpal tunnel syndrome (Nervous system disorders) | 19 (20) | 6 (6) | 7 (7)
Neuropathy peripheral (Nervous system disorders) | 16 (16) | 8 (8) | 7 (7)
Somnolence (Nervous system disorders) | 10 (10) | 10 (10) | 11 (11)
Tremor (Nervous system disorders) | 11 (11) | 5 (5) | 6 (6)
Cognitive disorder (Nervous system disorders) | 10 (10) | 5 (5) | 4 (4)
Dementia (Nervous system disorders) | 9 (9) | 5 (5) | 4 (4)
Sinus headache (Nervous system disorders) | 9 (9) | 2 (2) | 4 (5)
Amnesia (Nervous system disorders) | 7 (7) | 3 (3) | 4 (4)
Nerve compression (Nervous system disorders) | 5 (5) | 5 (5) | 4 (4)
Dysgeusia (Nervous system disorders) | 6 (6) | 4 (4) | 3 (3)
Tension headache (Nervous system disorders) | 8 (10) | 2 (2) | 3 (3)
Diabetic neuropathy (Nervous system disorders) | 7 (7) | 1 (1) | 3 (3)
Neuralgia (Nervous system disorders) | 6 (7) | 2 (2) | 3 (3)
Balance disorder (Nervous system disorders) | 4 (4) | 1 (1) | 5 (5)
Presyncope (Nervous system disorders) | 5 (5) | 3 (3) | 2 (2)
Restless legs syndrome (Nervous system disorders) | 5 (5) | 3 (3) | 2 (2)
Dementia Alzheimer's type (Nervous system disorders) | 3 (3) | 4 (4) | 2 (2)
Bell's palsy (Nervous system disorders) | 3 (3) | 3 (3) | 2 (2)
Parkinson's disease (Nervous system disorders) | 4 (4) | 2 (2) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 4 (4) | 2 (2) | 2 (2)
Memory impairment (Nervous system disorders) | 4 (4) | 1 (1) | 2 (2)
Brain fog (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3)
Head discomfort (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2)
Radiculopathy (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3)
Ageusia (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2)
Burning sensation (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2)
Cervical radiculopathy (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1)
Loss of consciousness (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Disturbance in attention (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Intercostal neuralgia (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Ophthalmic migraine (Nervous system disorders) | 0 (0) | 3 (4) | 1 (1)
Polyneuropathy (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Post-traumatic headache (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Anosmia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Cluster headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Essential tremor (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Parkinsonism (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Nervous system disorder (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Resting tremor (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Tardive dyskinesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Amnestic disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Apraxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Axonal and demyelinating polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Axonal neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Brain hypoxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebellar atrophy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral amyloid angiopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Coordination abnormal (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Crocodile tears syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dementia of the Alzheimer's type, uncomplicated (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Drooling (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dural arteriovenous fistula (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Facial spasm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Formication (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hyposmia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
IVth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Mental impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Micrographia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Motor dysfunction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Movement disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Occipital neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral nerve paresis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sensory disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sensory loss (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep deficit (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spasmodic dysphonia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal claudication (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Thunderclap headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Toxic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient global amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vestibular migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 299 (343) | 226 (245) | 261 (300)
Myalgia (Musculoskeletal and connective tissue disorders) | 205 (237) | 228 (249) | 307 (362)
Back pain (Musculoskeletal and connective tissue disorders) | 181 (195) | 87 (91) | 93 (100)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 98 (103) | 82 (89) | 91 (99)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 86 (86) | 49 (49) | 53 (57)
Neck pain (Musculoskeletal and connective tissue disorders) | 51 (52) | 25 (28) | 35 (36)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 33 (34) | 22 (22) | 23 (25)
Arthritis (Musculoskeletal and connective tissue disorders) | 26 (27) | 16 (17) | 12 (12)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 30 (30) | 13 (13) | 9 (9)
Bursitis (Musculoskeletal and connective tissue disorders) | 22 (22) | 11 (11) | 14 (14)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 15 (15) | 12 (13) | 18 (19)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 22 (22) | 10 (10) | 10 (10)
Osteopenia (Musculoskeletal and connective tissue disorders) | 17 (17) | 9 (9) | 8 (8)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 15 (16) | 11 (12) | 6 (6)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 12 (12) | 8 (9) | 10 (10)
Joint swelling (Musculoskeletal and connective tissue disorders) | 16 (16) | 8 (8) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 6 (6) | 10 (10)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 17 (17) | 8 (8) | 3 (3)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 14 (14) | 6 (6) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (6) | 5 (5)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 10 (11) | 4 (4) | 4 (4)
Trigger finger (Musculoskeletal and connective tissue disorders) | 8 (8) | 2 (2) | 7 (7)
Spinal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7) | 6 (6)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5) | 5 (5)
Foot deformity (Musculoskeletal and connective tissue disorders) | 9 (9) | 4 (4) | 2 (2)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 9 (9) | 4 (4) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (4) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 7 (7)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3) | 3 (3)
Exostosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 5 (5)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 8 (8) | 2 (2) | 2 (2)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 8 (8) | 2 (2) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (8) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 5 (5)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 4 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 2 (2)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 2 (2)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 2 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (2) | 3 (3)
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 2 (2)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 2 (2)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Costochondritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (3) | 0 (0)
Temporomandibular pain and dysfunction syndrome (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (2)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Sacroiliac joint dysfunction (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Clubbing (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Meniscopathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Palindromic rheumatism (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Articular calcification (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bone callus excessive (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bone loss (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Chondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Diffuse idiopathic skeletal hyperostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Enthesopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Exostosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Gouty tophus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Infrapatellar fat pad inflammation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc annular tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint lock (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ligament pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Limb deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Mastication disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteomalacia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Polychondritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Seronegative arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tarsi syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 229 (241) | 128 (139) | 135 (143)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 202 (225) | 141 (156) | 127 (133)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 194 (208) | 121 (127) | 88 (101)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 98 (108) | 51 (53) | 51 (53)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 71 (90) | 33 (38) | 37 (44)
Asthma (Respiratory, thoracic and mediastinal disorders) | 54 (62) | 31 (41) | 23 (27)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 53 (56) | 23 (23) | 29 (31)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 42 (44) | 30 (30) | 27 (27)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 42 (42) | 14 (15) | 30 (30)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 44 (46) | 25 (25) | 17 (18)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 29 (31) | 5 (5) | 13 (13)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 11 (12) | 16 (17)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 8 (8) | 10 (10)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 15 (15) | 6 (6)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 4 (4) | 4 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 6 (6) | 4 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 4 (4) | 4 (4)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 4 (4) | 4 (4)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 5 (6)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6) | 3 (3)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 7 (8) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 2 (2)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 3 (3)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 5 (5)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 2 (2)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 4 (4)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 2 (2) | 0 (0)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 0 (0)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchial wall thickening (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cystic lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lung hyperinflation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal cavity mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal crusting (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Neurogenic cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Paranasal sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal paraesthesia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinonasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Suffocation feeling (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Throat clearing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Throat lesion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tonsillar cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tracheal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 217 (230) | 119 (129) | 107 (110)
Nausea (Gastrointestinal disorders) | 70 (72) | 70 (73) | 76 (79)
Vomiting (Gastrointestinal disorders) | 51 (53) | 28 (30) | 27 (27)
Abdominal pain upper (Gastrointestinal disorders) | 47 (51) | 23 (23) | 29 (30)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 51 (51) | 13 (13) | 31 (31)
Abdominal pain (Gastrointestinal disorders) | 38 (41) | 24 (25) | 21 (21)
Toothache (Gastrointestinal disorders) | 35 (35) | 22 (24) | 19 (19)
Constipation (Gastrointestinal disorders) | 25 (28) | 22 (22) | 20 (21)
Dyspepsia (Gastrointestinal disorders) | 24 (24) | 12 (13) | 14 (15)
Gastritis (Gastrointestinal disorders) | 21 (21) | 9 (9) | 8 (8)
Dental caries (Gastrointestinal disorders) | 21 (22) | 2 (2) | 8 (8)
Large intestine polyp (Gastrointestinal disorders) | 14 (14) | 6 (7) | 11 (12)
Abdominal discomfort (Gastrointestinal disorders) | 13 (13) | 7 (7) | 8 (8)
Inguinal hernia (Gastrointestinal disorders) | 7 (7) | 8 (8) | 11 (11)
Umbilical hernia (Gastrointestinal disorders) | 10 (11) | 6 (6) | 5 (5)
Haemorrhoids (Gastrointestinal disorders) | 11 (11) | 2 (2) | 7 (7)
Dry mouth (Gastrointestinal disorders) | 11 (11) | 4 (5) | 4 (5)
Hiatus hernia (Gastrointestinal disorders) | 7 (7) | 5 (5) | 7 (7)
Dysphagia (Gastrointestinal disorders) | 7 (7) | 2 (2) | 5 (5)
Food poisoning (Gastrointestinal disorders) | 7 (7) | 2 (2) | 5 (5)
Abdominal pain lower (Gastrointestinal disorders) | 6 (6) | 3 (3) | 3 (3)
Irritable bowel syndrome (Gastrointestinal disorders) | 3 (4) | 5 (5) | 4 (4)
Mouth ulceration (Gastrointestinal disorders) | 5 (5) | 3 (3) | 2 (2)
Colitis (Gastrointestinal disorders) | 5 (5) | 2 (2) | 2 (2)
Diverticulum intestinal (Gastrointestinal disorders) | 3 (3) | 1 (1) | 5 (5)
Flatulence (Gastrointestinal disorders) | 5 (5) | 2 (2) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 6 (6) | 2 (2) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 5 (5) | 2 (2) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 4 (4) | 0 (0) | 2 (2)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Colitis microscopic (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3)
Colitis ulcerative (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4)
Gastrointestinal pain (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Odynophagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3)
Salivary hypersecretion (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 3 (5) | 2 (2) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Faeces soft (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Glossodynia (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Enteritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Melaena (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Pancreatic failure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Peptic ulcer (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Bile acid malabsorption (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Coeliac disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Epiploic appendagitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal tract irritation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gingival disorder (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Glossitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Lip pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Noninfective gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Rectal tenesmus (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal symptom (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anal eczema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Angular cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Appendix disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulum oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenogastric reflux (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival recession (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gingival ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lip disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mesenteric artery stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral mucosal exfoliation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral papule (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatic disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatic steatosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Parotid gland enlargement (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Precancerous lesion of digestive tract (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Proctitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyloric sphincter insufficiency (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Reflux gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Salivary duct obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Salivary gland pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Steatorrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tongue coated (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tongue dry (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth deposit (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 54 (55) | 28 (28) | 30 (30)
Contusion (Injury, poisoning and procedural complications) | 45 (46) | 22 (23) | 14 (14)
Arthropod bite (Injury, poisoning and procedural complications) | 23 (24) | 16 (16) | 21 (22)
Skin laceration (Injury, poisoning and procedural complications) | 29 (30) | 16 (16) | 10 (10)
Ligament sprain (Injury, poisoning and procedural complications) | 25 (25) | 15 (16) | 9 (9)
Limb injury (Injury, poisoning and procedural complications) | 17 (17) | 17 (18) | 11 (11)
Muscle strain (Injury, poisoning and procedural complications) | 24 (25) | 10 (10) | 11 (11)
Procedural pain (Injury, poisoning and procedural complications) | 21 (22) | 12 (12) | 7 (7)
Tooth fracture (Injury, poisoning and procedural complications) | 21 (21) | 5 (5) | 9 (9)
Foot fracture (Injury, poisoning and procedural complications) | 16 (16) | 9 (9) | 5 (5)
Immunisation reaction (Injury, poisoning and procedural complications) | 13 (14) | 4 (4) | 9 (9)
Rib fracture (Injury, poisoning and procedural complications) | 16 (16) | 5 (5) | 5 (6)
Arthropod sting (Injury, poisoning and procedural complications) | 13 (15) | 4 (4) | 6 (6)
Joint injury (Injury, poisoning and procedural complications) | 16 (16) | 3 (3) | 3 (3)
Head injury (Injury, poisoning and procedural complications) | 9 (9) | 5 (5) | 7 (7)
Wrist fracture (Injury, poisoning and procedural complications) | 8 (8) | 5 (5) | 8 (8)
Animal bite (Injury, poisoning and procedural complications) | 9 (9) | 6 (6) | 3 (3)
Meniscus injury (Injury, poisoning and procedural complications) | 9 (9) | 5 (5) | 4 (4)
Soft tissue injury (Injury, poisoning and procedural complications) | 10 (10) | 5 (5) | 3 (3)
Hand fracture (Injury, poisoning and procedural complications) | 10 (10) | 2 (2) | 4 (4)
Radius fracture (Injury, poisoning and procedural complications) | 6 (6) | 7 (7) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 9 (10) | 3 (3) | 3 (3)
Tendon rupture (Injury, poisoning and procedural complications) | 7 (7) | 5 (5) | 3 (4)
Ligament rupture (Injury, poisoning and procedural complications) | 5 (5) | 5 (5) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 8 (8) | 1 (1) | 3 (3)
Clavicle fracture (Injury, poisoning and procedural complications) | 8 (8) | 0 (0) | 3 (3)
Craniofacial fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 7 (7)
Ankle fracture (Injury, poisoning and procedural complications) | 4 (4) | 3 (3) | 3 (3)
Bone contusion (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 4 (4)
Fibula fracture (Injury, poisoning and procedural complications) | 4 (4) | 4 (4) | 2 (2)
Concussion (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 4 (4)
Lower limb fracture (Injury, poisoning and procedural complications) | 7 (7) | 1 (1) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 5 (5) | 2 (2) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 4 (4)
Eye injury (Injury, poisoning and procedural complications) | 6 (6) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 4 (4) | 3 (3) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 5 (6) | 2 (2) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 5 (5) | 2 (2) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 3 (3)
Chest injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 2 (2)
Epicondylitis (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 3 (3)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 5 (5) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 2 (2)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 2 (2)
Back injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1)
Exposure to SARS-CoV-2 (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Wound (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Musculoskeletal foreign body (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Synovial rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Foreign body in throat (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Fractured coccyx (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Heat illness (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Hypobarism (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Muscle contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Post procedural contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Radiation injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Avulsion fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Bone fragmentation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Burn oral cavity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Chemical burns of eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Chillblains (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Corneal epithelial downgrowth (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Dental restoration failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Electric shock (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Foreign body in ear (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hyphaema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Injection related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Metal poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Neck injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Open fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Penis injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Renal transplant failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Snake bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Sports injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Venomous sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 246 (250) | 110 (111) | 107 (110)
Hypotension (Vascular disorders) | 19 (20) | 9 (10) | 7 (7)
Haematoma (Vascular disorders) | 14 (14) | 2 (2) | 5 (5)
Hot flush (Vascular disorders) | 7 (7) | 8 (8) | 5 (5)
Deep vein thrombosis (Vascular disorders) | 8 (8) | 6 (6) | 4 (4)
Peripheral arterial occlusive disease (Vascular disorders) | 6 (6) | 4 (5) | 2 (2)
Peripheral vascular disorder (Vascular disorders) | 7 (7) | 2 (2) | 2 (2)
Peripheral venous disease (Vascular disorders) | 7 (7) | 2 (2) | 2 (2)
Varicose vein (Vascular disorders) | 7 (7) | 1 (1) | 1 (1)
Thrombosis (Vascular disorders) | 4 (4) | 1 (1) | 2 (2)
Aortic aneurysm (Vascular disorders) | 3 (3) | 2 (2) | 1 (1)
Aortic arteriosclerosis (Vascular disorders) | 2 (2) | 2 (2) | 2 (2)
Aortic stenosis (Vascular disorders) | 3 (4) | 2 (2) | 1 (1)
Flushing (Vascular disorders) | 1 (2) | 1 (1) | 4 (4)
Hypertensive crisis (Vascular disorders) | 2 (2) | 1 (1) | 3 (3)
Phlebitis (Vascular disorders) | 3 (3) | 1 (1) | 2 (2)
Lymphoedema (Vascular disorders) | 3 (3) | 0 (0) | 2 (3)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 3 (3) | 0 (0)
Thrombophlebitis (Vascular disorders) | 3 (3) | 1 (1) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 3 (3)
Blood pressure fluctuation (Vascular disorders) | 2 (2) | 2 (2) | 0 (0)
Essential hypertension (Vascular disorders) | 2 (2) | 0 (0) | 2 (2)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (1) | 3 (3)
Giant cell arteritis (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
White coat hypertension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Aortic dilatation (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Intermittent claudication (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Peripheral artery occlusion (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Aortic disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Bleeding varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Blood pressure inadequately controlled (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Microscopic polyangiitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Phlebectasia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Phlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Subclavian steal syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Systolic hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Varicose ulceration (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vasodilatation (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 55 (56) | 22 (22) | 39 (39)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 60 (60) | 24 (25) | 20 (20)
Gout (Metabolism and nutrition disorders) | 36 (38) | 19 (20) | 20 (23)
Hyperlipidaemia (Metabolism and nutrition disorders) | 39 (39) | 13 (13) | 16 (16)
Decreased appetite (Metabolism and nutrition disorders) | 24 (24) | 19 (19) | 21 (22)
Vitamin D deficiency (Metabolism and nutrition disorders) | 21 (21) | 12 (12) | 18 (18)
Diabetes mellitus (Metabolism and nutrition disorders) | 20 (20) | 15 (16) | 11 (11)
Dyslipidaemia (Metabolism and nutrition disorders) | 20 (20) | 6 (6) | 6 (6)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 17 (17) | 7 (7) | 8 (8)
Hyperuricaemia (Metabolism and nutrition disorders) | 9 (9) | 6 (6) | 7 (7)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 8 (8) | 4 (4) | 8 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 9 (9) | 3 (3) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (6) | 5 (5) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (7) | 4 (4) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 3 (3) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 4 (4) | 5 (5) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 2 (2)
Iron deficiency (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (5)
Impaired fasting glucose (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Insulin resistance (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Calcium deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Enzyme abnormality (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Gluten sensitivity (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypovitaminosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Lipoedema (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Magnesium deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Overweight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Vitamin B1 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Vitamin B6 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 36 (36) | 31 (31) | 36 (36)
Pruritus (Skin and subcutaneous tissue disorders) | 34 (34) | 24 (25) | 17 (17)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 21 (21) | 12 (13) | 13 (13)
Erythema (Skin and subcutaneous tissue disorders) | 17 (17) | 6 (6) | 13 (13)
Urticaria (Skin and subcutaneous tissue disorders) | 13 (13) | 14 (15) | 7 (8)
Eczema (Skin and subcutaneous tissue disorders) | 15 (16) | 9 (9) | 8 (8)
Skin lesion (Skin and subcutaneous tissue disorders) | 7 (7) | 12 (14) | 8 (10)
Dermatitis (Skin and subcutaneous tissue disorders) | 12 (12) | 4 (4) | 7 (7)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 11 (12) | 7 (7) | 4 (4)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 13 (14) | 1 (1) | 4 (4)
Skin ulcer (Skin and subcutaneous tissue disorders) | 8 (9) | 2 (2) | 7 (7)
Psoriasis (Skin and subcutaneous tissue disorders) | 7 (7) | 3 (3) | 6 (6)
Night sweats (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5) | 6 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6) | 3 (3)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 8 (8) | 1 (1) | 4 (4)
Rash pruritic (Skin and subcutaneous tissue disorders) | 3 (6) | 5 (5) | 2 (2)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 2 (2)
Dermal cyst (Skin and subcutaneous tissue disorders) | 6 (7) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Lichen planus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Skin warm (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Blood blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Granuloma annulare (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Sensitive skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Alopecia scarring (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Androgenetic alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Keloid scar (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lentigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lichen planopilaris (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Milia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myxoid cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Onychogryphosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pemphigus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Photodermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Purpura senile (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sebaceous gland disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin lesion inflammation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spider naevus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 90 (96) | 35 (36) | 32 (33)
Palpitations (Cardiac disorders) | 20 (22) | 10 (11) | 5 (5)
Angina pectoris (Cardiac disorders) | 11 (11) | 5 (6) | 10 (12)
Tachycardia (Cardiac disorders) | 12 (12) | 9 (9) | 3 (3)
Bradycardia (Cardiac disorders) | 10 (10) | 4 (4) | 8 (8)
Coronary artery disease (Cardiac disorders) | 6 (6) | 6 (6) | 7 (7)
Cardiac failure congestive (Cardiac disorders) | 7 (7) | 6 (6) | 5 (5)
Arrhythmia (Cardiac disorders) | 9 (9) | 4 (4) | 4 (4)
Cardiac failure (Cardiac disorders) | 9 (9) | 2 (2) | 5 (5)
Myocardial ischaemia (Cardiac disorders) | 6 (6) | 3 (3) | 3 (3)
Extrasystoles (Cardiac disorders) | 7 (7) | 2 (2) | 0 (0)
Atrial flutter (Cardiac disorders) | 2 (2) | 5 (5) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 2 (2) | 3 (3) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 5 (5) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 3 (3) | 1 (1) | 2 (2)
Cardiac failure chronic (Cardiac disorders) | 4 (4) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 3 (3) | 2 (2) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Bundle branch block right (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Cardiomegaly (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Tachycardia paroxysmal (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Chronic coronary syndrome (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Heart failure with reduced ejection fraction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Heart valve incompetence (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Mitral valve calcification (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Mitral valve prolapse (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Aortic valve calcification (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bundle branch block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Dilated cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myopericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Right ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinoatrial block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 56 (63) | 19 (20) | 22 (23)
Eye pain (Eye disorders) | 11 (11) | 8 (8) | 9 (9)
Glaucoma (Eye disorders) | 17 (17) | 3 (3) | 8 (10)
Dry eye (Eye disorders) | 14 (14) | 4 (4) | 7 (7)
Lacrimation increased (Eye disorders) | 13 (15) | 6 (6) | 6 (6)
Macular degeneration (Eye disorders) | 6 (6) | 10 (10) | 5 (5)
Eye pruritus (Eye disorders) | 10 (10) | 4 (4) | 1 (1)
Blepharitis (Eye disorders) | 4 (4) | 6 (7) | 2 (2)
Vision blurred (Eye disorders) | 5 (5) | 3 (3) | 2 (2)
Retinal detachment (Eye disorders) | 4 (4) | 3 (3) | 1 (1)
Vitreous detachment (Eye disorders) | 3 (3) | 2 (2) | 2 (2)
Conjunctival haemorrhage (Eye disorders) | 3 (3) | 1 (1) | 2 (2)
Ocular hyperaemia (Eye disorders) | 6 (6) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 3 (4) | 2 (2) | 1 (1)
Visual impairment (Eye disorders) | 1 (1) | 1 (1) | 4 (4)
Conjunctivitis allergic (Eye disorders) | 4 (4) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 2 (2) | 1 (1) | 2 (2)
Eye irritation (Eye disorders) | 3 (3) | 1 (1) | 1 (1)
Diplopia (Eye disorders) | 4 (5) | 0 (0) | 0 (0)
Epiretinal membrane (Eye disorders) | 2 (2) | 1 (1) | 1 (1)
Eye disorder (Eye disorders) | 2 (2) | 1 (1) | 1 (1)
Eye swelling (Eye disorders) | 2 (2) | 1 (1) | 1 (1)
Vitreous floaters (Eye disorders) | 3 (3) | 0 (0) | 1 (1)
Asthenopia (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 3 (3) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 2 (2) | 0 (0) | 1 (1)
Macular hole (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
Neovascular age-related macular degeneration (Eye disorders) | 2 (2) | 0 (0) | 1 (1)
Posterior capsule opacification (Eye disorders) | 0 (0) | 3 (3) | 0 (0)
Retinal artery occlusion (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Swelling of eyelid (Eye disorders) | 1 (1) | 0 (0) | 2 (2)
Dacryostenosis acquired (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Entropion (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Eye allergy (Eye disorders) | 1 (1) | 1 (3) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Eyelid cyst (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Eyelid pain (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Keratitis (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Abnormal sensation in eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract nuclear (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Choroidal neovascularisation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatochalasis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dry age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema eyelids (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema of eyelid (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye degenerative disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye haematoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye inflammation (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye ulcer (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eyelid margin crusting (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid skin dryness (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelids pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Iridocyclitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Lacrimal fistula (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Macular scar (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Maculopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Meibomian gland dysfunction (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Metamorphopsia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Narrow anterior chamber angle (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Ocular discomfort (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ocular hypertension (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Optic nerve sheath haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Periorbital swelling (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Pinguecula (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Pterygium (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal infarction (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal neovascularisation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal vascular thrombosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinopathy hypertensive (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Scleral hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Scleritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Trichiasis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Visual field defect (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vitreous opacities (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 5 (6) | 15 (15) | 39 (42)
Blood pressure increased (Investigations) | 31 (31) | 13 (13) | 10 (10)
SARS-CoV-2 test positive (Investigations) | 17 (17) | 9 (9) | 11 (12)
Weight decreased (Investigations) | 9 (9) | 9 (9) | 4 (4)
Blood cholesterol increased (Investigations) | 8 (8) | 4 (4) | 8 (8)
Cardiac murmur (Investigations) | 6 (6) | 7 (7) | 5 (5)
Prostatic specific antigen increased (Investigations) | 7 (7) | 3 (3) | 3 (3)
Heart rate increased (Investigations) | 5 (5) | 4 (4) | 2 (2)
Heart rate irregular (Investigations) | 5 (5) | 2 (2) | 1 (1)
Blood glucose increased (Investigations) | 2 (2) | 3 (3) | 1 (1)
Weight increased (Investigations) | 3 (3) | 0 (0) | 3 (3)
Blood creatinine increased (Investigations) | 5 (5) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 2 (2) | 2 (2) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 2 (2) | 2 (2) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (2) | 3 (3) | 0 (0)
Blood pressure decreased (Investigations) | 3 (3) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 4 (4) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Blood testosterone decreased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Chest X-ray abnormal (Investigations) | 1 (1) | 1 (1) | 1 (1)
Intraocular pressure increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Blood glucose decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood pressure abnormal (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Bone density decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Helicobacter test positive (Investigations) | 1 (1) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Occult blood positive (Investigations) | 1 (1) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Rheumatoid factor increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
SARS-CoV-2 antibody test positive (Investigations) | 2 (2) | 0 (0) | 0 (0)
Serum ferritin decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Urine output increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Vitamin B12 decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Allergy test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Antinuclear antibody positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Biopsy (Investigations) | 0 (0) | 0 (0) | 1 (1)
Biopsy breast (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood glucose abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood immunoglobulin E increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood immunoglobulin G decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood iron increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood pressure diastolic increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Body temperature decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Brain natriuretic peptide increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Breast scan abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Carcinoembryonic antigen increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Colonoscopy (Investigations) | 0 (0) | 0 (0) | 1 (1)
Computerised tomogram thorax abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cystoscopy (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electroencephalogram abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
HIV test positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis B surface antibody positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Influenza B virus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Investigation abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lipids abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Occult blood (Investigations) | 0 (0) | 0 (0) | 1 (1)
Pulse abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Respiratory rate increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Sputum abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Total lung capacity decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21 (21) | 21 (23) | 15 (15)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 (19) | 11 (11) | 7 (7)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 6 (6) | 3 (3)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 5 (5) | 4 (4)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 3 (3) | 4 (4)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 0 (0) | 2 (2)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (3) | 2 (2)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4) | 2 (2)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1) | 3 (3)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 3 (3)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 2 (2)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Benign soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Adenoid cystic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
B-cell type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Benign hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia stage 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ear neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
High-grade B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lipoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Mucinous breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ocular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal hamartoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Skull base tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Small cell lung cancer limited stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Splenic marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Urethral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 52 (52) | 18 (18) | 20 (20)
Insomnia (Psychiatric disorders) | 37 (37) | 21 (21) | 23 (24)
Anxiety (Psychiatric disorders) | 19 (19) | 25 (25) | 23 (25)
Sleep disorder (Psychiatric disorders) | 4 (4) | 4 (4) | 5 (5)
Stress (Psychiatric disorders) | 5 (5) | 1 (1) | 2 (2)
Confusional state (Psychiatric disorders) | 2 (2) | 3 (3) | 1 (1)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 3 (3) | 0 (0) | 2 (2)
Restlessness (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1)
Panic attack (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1)
Alcoholism (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Nightmare (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Persistent depressive disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Apathy (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Middle insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Mood swings (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Obsessive-compulsive disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Poor quality sleep (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Agoraphobia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anger (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anhedonia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Binge eating (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Emotional disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Grief reaction (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Habit cough (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Neurosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Panic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep terror (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Somnambulism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Terminal insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 47 (52) | 26 (26) | 20 (20)
Ear pain (Ear and labyrinth disorders) | 30 (31) | 13 (13) | 16 (17)
Tinnitus (Ear and labyrinth disorders) | 20 (21) | 7 (8) | 9 (9)
Vertigo positional (Ear and labyrinth disorders) | 7 (8) | 1 (1) | 3 (3)
Cerumen impaction (Ear and labyrinth disorders) | 7 (7) | 2 (2) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 5 (5) | 0 (0) | 5 (5)
Hypoacusis (Ear and labyrinth disorders) | 4 (5) | 1 (1) | 3 (3)
Deafness (Ear and labyrinth disorders) | 4 (4) | 1 (1) | 1 (1)
Deafness bilateral (Ear and labyrinth disorders) | 2 (2) | 3 (3) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 2 (2)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 2 (2)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 3 (3) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 1 (1)
Ear congestion (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Ear inflammation (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Inner ear disorder (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Motion sickness (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Otosclerosis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Tympanic membrane disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Deafness transitory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Ear haemorrhage (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Eustachian tube obstruction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Inner ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 16 (16) | 10 (10) | 7 (7)
Hypertonic bladder (Renal and urinary disorders) | 13 (13) | 8 (8) | 5 (5)
Haematuria (Renal and urinary disorders) | 10 (10) | 4 (4) | 5 (5)
Pollakiuria (Renal and urinary disorders) | 7 (7) | 2 (2) | 9 (9)
Urinary incontinence (Renal and urinary disorders) | 8 (8) | 3 (3) | 7 (7)
Chronic kidney disease (Renal and urinary disorders) | 8 (8) | 7 (7) | 2 (2)
Dysuria (Renal and urinary disorders) | 8 (8) | 5 (5) | 3 (3)
Renal cyst (Renal and urinary disorders) | 3 (3) | 7 (7) | 6 (6)
Urinary retention (Renal and urinary disorders) | 7 (7) | 3 (3) | 6 (6)
Renal failure (Renal and urinary disorders) | 7 (7) | 0 (0) | 2 (2)
Urinary tract inflammation (Renal and urinary disorders) | 3 (4) | 1 (1) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 2 (2) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 1 (1) | 3 (3)
Renal colic (Renal and urinary disorders) | 4 (5) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 3 (4) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Bladder dysfunction (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Cystitis interstitial (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Lower urinary tract symptoms (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Nephropathy (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Renal atrophy (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Renal disorder (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Urinary tract disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotonic urinary bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ketonuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Microalbuminuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal cyst haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal cyst ruptured (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urethral disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Vesical fistula (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 33 (33) | 8 (8) | 21 (21)
Prostatomegaly (Reproductive system and breast disorders) | 7 (7) | 1 (1) | 6 (6)
Prostatitis (Reproductive system and breast disorders) | 5 (5) | 4 (4) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 4 (4) | 3 (3) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 2 (2) | 5 (5) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 5 (5) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 3 (3) | 1 (1)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 2 (2)
Uterine prolapse (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 (3) | 1 (1) | 0 (0)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 1 (2) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Prostatic mass (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
Testicular swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Bartholin's cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Breast discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2)
Coital bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Endometrial thickening (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Epididymal cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Genital haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Macroorchidism (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Perineal rash (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatic disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Rectocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Scrotal swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 24 (24) | 14 (14) | 10 (10)
Lymphadenopathy (Blood and lymphatic system disorders) | 10 (11) | 11 (11) | 13 (15)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 18 (18) | 4 (4) | 6 (6)
Lymph node pain (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1)
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Pernicious anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Anaemia folate deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Bone marrow oedema (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Macrocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Spleen disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
White blood cell disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 19 (19) | 16 (16) | 20 (21)
Drug hypersensitivity (Immune system disorders) | 3 (3) | 3 (3) | 6 (6)
Hypersensitivity (Immune system disorders) | 5 (5) | 2 (2) | 3 (3)
Multiple allergies (Immune system disorders) | 2 (2) | 1 (1) | 3 (3)
Food allergy (Immune system disorders) | 3 (3) | 0 (0) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 2 (2) | 0 (0) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Allergy to chemicals (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Allergy to vaccine (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Dust allergy (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Allergy to plants (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Amyloidosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Mycotic allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Rubber sensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 24 (25) | 10 (10) | 9 (9)
Hyperthyroidism (Endocrine disorders) | 7 (7) | 2 (2) | 2 (2)
Thyroid mass (Endocrine disorders) | 7 (7) | 2 (2) | 2 (2)
Goitre (Endocrine disorders) | 6 (6) | 1 (1) | 1 (1)
Hypogonadism (Endocrine disorders) | 2 (2) | 2 (2) | 1 (1)
Graves' disease (Endocrine disorders) | 3 (3) | 0 (0) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 2 (2) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 2 (2) | 0 (0)
Adrenal mass (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Autoimmune hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Primary hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Thyroid cyst (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Toxic nodular goitre (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 12 (12) | 1 (1) | 4 (4)
Hepatic steatosis (Hepatobiliary disorders) | 6 (6) | 3 (3) | 6 (6)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 1 (1)
Hepatic mass (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Non-alcoholic fatty liver (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Type V hyperlipidaemia (Congenital, familial and genetic disorders) | 1 (1) | 1 (1) | 0 (0)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Epidermal naevus (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Frenulum breve (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Porokeratosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth hypoplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Turner's syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Device breakage (Product Issues) | 2 (2) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Ex-tobacco user (Social circumstances) | 0 (0) | 0 (0) | 1 (1)
Immobile (Social circumstances) | 0 (0) | 0 (0) | 1 (1)
Menopause (Social circumstances) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT04886596/Prot_003.pdf
  • Statistical Analysis Plan (2024-06-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT04886596/SAP_004.pdf